## MC1973 / 19-011871

A Phase II Study of Hypofractionated Pre-Operative Radiation Therapy for Localized, Resectable Soft Tissue Sarcoma of the Extremity or Superficial Trunk

NCT04562480

Document Date: 04/17/2024

## Mayo Clinic: Department of Radiation Oncology

# MC1973: A Phase II Study of Hypofractionated Pre-Operative Radiation Therapy for Localized, Resectable Soft Tissue Sarcoma of the Extremity and Superficial Trunk

Study Chair: Safia Ahmed, M.D.

Mayo Clinic

Department of Radiation Oncology

5777 E. Mayo Blvd Phoenix, AZ, 85054

Study Co-Investigators: Ivy Petersen, M.D.

Matthew T. Houdek, M.D.

Peter S. Rose, M.D. Brittany L. Siontis, M.D. James L. Leenstra, M.D.

Michael Rutenberg, M.D., Ph.D. Meng Welliver, M.D., Ph.D.

Statisticians: Maddy Dorr, M.S.√

Study Contributor(s): Yeoniee Kim, B.S.  $\sqrt{}$ 

√Study contributor(s) not responsible for patient care

## **Document History**

| Version 1 | 5/20/2020 |
|-----------|------------|
| Version 2 | 10/16/2020 |
| Version 3 | 12/09/2020 |
| Version 4 | 01/22/2021 |
| Version 5 | 03/30/2021 |
| Version 6 | 03/04/2022 |

| Version 7 | 7/18/2022 |
|------------|-----------|
| Version 8 | 2/20/2023 |
| Version 9 | 5/4/2023 |
| Version 10 | 7/20/2023 |
| Version 11 | 9/05/2023 |
| Version 12 | 1/04/2024 |
| Version 13 | 4/17/2024 |

## **Protocol Resources**

| Questions: | Contact Name: |
|---|---|
| Patient eligibility, test schedule, treatment delays/interruptions/ adjustments, dose modifications, forms completion/ submission, & adverse events | Radiation Oncology Study Team Contacts listed on the consent form |
| Protocol document, consent form and regulatory issues | Yeoniee Kim. B.S.<br>E-mail: kim.yeoniee@mayo.edu |
| Statisticians | Maddy Dorr, M.S.<br>E-mail: dorr.madeline@mayo.edu |

## **Table of Contents**

| Protoco | ol Resources | 2 |
|---------|-------------------------------------------------------|----|
| Table o | of Contents | 3 |
| Study S | Schema | 4 |
| List of | Abbreviations | 5 |
| 1.0 | Background and Rationale | 6 |
| 2.0 | Goals | 8 |
| 3.0 | Patient Eligibility | 8 |
| 4.0 | Test Schedule | 11 |
| 5.0 | Stratification Factors OR Grouping Factor | 11 |
| 6.0 | Registration/Procedures | 11 |
| 7.0 | Protocol Treatment | 11 |
| 8.0 | Dosage Modification Based on Adverse Events | 19 |
| 9.0 | Ancillary Treatment/Supportive Care | 19 |
| 10.0 | Adverse Event (AE) Monitoring and Reporting | 19 |
| 11.0 | Treatment Evaluation/Measurement of Effect | 25 |
| 12.0 | Descriptive Factors | 25 |
| 13.0 | Treatment/Follow-up Decision at Evaluation of Patient | 26 |
| 14.0 | Body Fluid Biospecimens | 27 |
| 15.0 | Drug Information. | 27 |
| 16.0 | Statistical Considerations and Methodology | 27 |
| 17.0 | Pathology Considerations/Tissue Biospecimens | 34 |
| 18.0 | Records and Data Collection Procedures | 34 |
| 19.0 | Budget | 34 |
| 20.0 | References | 35 |
| Append | dix I ECOG Performance Status | 37 |
| Append | dix II PROMIS | 48 |
| Append | dix III TESS | 49 |
| Append | dix IV Joint Stiffness Assessment | 72 |
| Append | dix V Regional Alopecia Assessment | 73 |
| Annend | dix VI Surgical Wound Complication Assessment | 7 |

3

## **Study Schema**

Localized, resectable soft tissue sarcoma of the extremity/limb girdle or superficial trunk

 $\downarrow$ 

Pre-operative radiation therapy

Dose: 42.75 Gy in 15 fractions

 $\downarrow$ 

Definitive surgical resection

(3-6 weeks interval between radiation therapy and definitive surgery)



**Event Monitoring** 

## **List of Abbreviations**

| AE | Adverse Event/Adverse Experience |
|---|---|
| BID | Twice daily |
| cGy | centiGray |
| CRF | Case Report Form |
| CT | Computed Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTV | Clinical Target Volume |
| DSMB | Data and Safety Monitoring Board |
| DVH | Dose Volume Histogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| ER / ES | Electronic Record and Electronic Signature |
| Gy | Gray |
| GTV | Gross Tumor Volume |
| ICRU | International Commission on Radiation Units and Measurements |
| IMPT | Intensity Modulated Proton Therapy |
| IMRT | Intensity Modulated Radiotherapy |
| IND / IDE | Investigational Drugs and Devices |
| IRB | Institutional Review Board |
| ITV | Internal Target Volume |
| LFR5 | Local Failure Rate at 5 years |
| MCCC | Mayo Clinic Cancer Center |
| MRI | Magnetic Resonance Imaging |
| PROMISE | Patient-Reported Outcomes Measurement Information System |
| PS | Performance Status |
| PTV | Planning Target Volume |
| RBE | Relative Biological Effectiveness |
| RT | Radiation Therapy |
| SOC | System Organ Class |
| TESS | Toronto Extremity Salvage Score |
| UPIRTSO | Unanticipated Problems Involving Risks To Subjects or Others |
| VMAT | Volumetric Modulated Arc Therapy |
| 3DCRT | 3D Conformal Radiation Therapy |

## 1.0 Background and Rationale

Approximately 12,000 patients are diagnosed with soft tissue sarcomas annually in the United States, accounting for 1% of all adult malignancies. Given the rarity, diversity (> 60 different histologies), and treatment complexity associated with soft tissue sarcomas, patients routinely undergo treatment at specialty centers. Historically, extremity soft tissue sarcomas were treated with amputation. Advances in radiation therapy and surgical techniques, however, have made radiation therapy plus limb-salvage surgery the standard treatment for most localized, extremity soft tissue sarcomas. Superficial trunk soft tissue sarcomas are treated in a similar fashion. With this multi-modal treatment approach, the 5 year local recurrence rate for extremity and superficial trunk soft tissue sarcomas is  $\leq 10\%$ .

Radiation therapy can be administered preoperatively, intraoperatively, postoperatively, or as a combination of the aforementioned.<sup>2,3,7</sup> Preoperative radiation therapy is associated with a higher acute wound complication rate compared to postoperative radiation therapy.<sup>6</sup> O'Sullivan et. al. reported a 35% acute wound complication rate with preoperative radiation therapy compared to a 17% rate with postoperative radiation.<sup>6</sup> Acute wound complication was defined as a major wound issue requiring an invasive intervention (i.e., second surgery or hospitalization for wound care) within 3 months of surgery.<sup>6</sup> Several other reports document similar acute wound complication rates.<sup>8-12</sup>

Many centers in the Unites States and abroad favor pre-operative radiation therapy due to the lower total radiation dose administered (50 Gray (Gy) versus 60-66 Gy) and smaller treatment volume compared to postoperative radiation therapy. These aspects are thought to contribute to the lower irreversible, long-term toxicity rates seen with preoperative radiation therapy. <sup>13,14</sup> Davis et. al. reported more frequent rates of fibrosis (48.2% versus 31.5%), edema (23.2% versus 15.1%), and joint stiffness (23.2% versus 17.8%) with postoperative radiation therapy compared to preoperative radiation therapy. <sup>14</sup> Higher rates of irreversible, long-term toxicities adversely affect patient function. <sup>13,14</sup> Lastly, preoperative radiation therapy optimizes the chances of obtaining a margin-negative resection and may decrease the potential for metastatic cell spread at time of surgery. <sup>6,8,15</sup>

The radiation therapy course for soft tissue sarcomas is certainly long, with total number of fractions ranging from 25 fractions (preoperative treatment) to 33 fractions (postoperative treatment). Given the financial and time commitments associated with the radiation treatment length, there are potential benefits for patients by reducing the number of daily fractions administered. Shorter treatment duration can translate to reduced costs and improved patient experiences due to reduced travel times, decreased time off work and away from family, and lessened financial demands associated with pursuing treatment at a specialty center. Additionally, a shorter radiation course may lead to higher limb preservation rates and improved survival in minority groups as outcomes are known to be inferior in African American and Latino populations compared to the Caucasian population. 16,17

One method to shorten radiation treatment length is to administer a hypofractionated treatment course. Hypofractionated radiation therapy administers the total radiation dose

as larger daily doses compared to conventionally fractionated therapy. This effectively reduces the overall treatment duration by weeks. Hypofractionated radiation therapy is proven to be a more convenient and lower cost option for early stage breast and prostate cancers, without compromising oncologic outcomes or increasing the likelihood of treatment-related side effects. <sup>18-20</sup> For example, Whelan et. al. demonstrated the efficacy of a hypofractionated postoperative treatment course (42.56 Gy in 16 fractions) for early stage breast cancer compared to conventionally fractionated treatment (50 Gy in 25 fractions). <sup>20</sup> At 10 years, the local recurrence rate was 6.7% for conventionally fractionated radiation therapy versus 6.7% for hypofractionated radiation therapy. <sup>20</sup> Additionally, there was no difference in overall survival or cosmetic outcomes between the two treatment arms. <sup>20</sup>

Hypofractionated radiation therapy has been studied to a more limited degree in soft tissue sarcomas. In Poland, a study of hypofractionated preoperative radiation therapy (25 Gy in 5 fractions) was conducted in 272 patients from 2006 to 2011.<sup>21</sup> This study yielded a higher local failure rate: 19%, with a median follow up of 35 months.<sup>21</sup> Of note, the biologic effective dose is 34.27 Gy<sub>10</sub> with this regimen compared to 43.83 Gy<sub>10</sub> with conventional fractionation, suggesting a higher biologic effective dose is needed with hypofractionation to achieve optimal outcomes. Another preoperative hypofractionated study from University of California Los Angeles studied 28 Gy in 8 fractions (biologic effective dose of 32.63 Gy). The local failure rate at 3 years was 11%. Again, these

results suggest a higher total radiation dose is needed for efficacy when utilizing a hypofractionated radiation treatment course in soft tissue sarcomas.

We propose conducting a single arm, prospective study to evaluate the efficacy and safety of a preoperative hypofractionated course, 42.75 Gy in 15 fractions, for localized, extremity and superficial trunk soft tissue sarcomas. The biologic equivalent dose of this regimen is 45.20 Gy<sub>10</sub>, similar to 43.83 Gy<sub>10</sub> associated with conventionally fractionated 50 Gy in 25 fractions. The primary aim of the study is to determine acute wound complications rates, as defined by O'Sullivan et. al.<sup>6</sup> Secondary aims will analyze local failure rate, disease-free survival, overall survival, patterns of relapse, late toxicities, and quality of life/patient-reported outcomes. We hypothesize a 15 fraction hypofractionated radiation therapy course will be associated with equivalent short-term toxicity rates and oncologic outcomes as compared to historical standards.

#### 2.0 Goals

## 2.1 Primary Objective

2.1.1 To report the major acute wound complication rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions. See section 11.1 for definition of major acute wound complications.

## 2.2 Secondary Objectives

- 2.2.1 To report the 5-year local failure rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.
- 2.2.2 To report the 5-year disease-free survival rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.
- 2.2.3 To report the 5-year overall survival rate associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.
- 2.2.4 To report long-term toxicity rates associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.
- 2.2.5 To describe patterns of relapse associated with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.
- 2.2.6 To describe patient reported outcomes/quality-of-life outcomes with hypofractionated preoperative radiation therapy, 42.75 Gy in 15 fractions.

## 3.0 Patient Eligibility

The patient must meet all selection criteria as specified in Section 3.1 and be agreeable to adhere to the follow-up evaluations and schedule. Written informed consent must be obtained from the patient prior to enrollment and prior to any trial-specific evaluations.

#### 3.1 Inclusion Criteria

- 3.1.1 Males and females age  $\geq$  18 years.
- 3.1.2 Newly diagnosed, histological confirmation of soft tissue sarcoma of the extremities (including limb girdle) or superficial trunk that present as either
  - Deemed a candidate for complete macroscopic resection of the primary sarcoma.

- Having had non-oncologic excisional procedure with positive or uncertain resection margins and still be eligible if the evaluating sarcoma surgeon recommends oncologic re-resection of the surgical bed to obtain negative margins after a course of preoperative radiation therapy.
- 3.1.3 No evidence of nodal or distant metastases as determined by clinical examination on any form of imaging.
- 3.1.4 Eastern Cooperative oncology Group (ECOG) Performance Status (PS)  $\leq$  3 (Appendix I).
- 3.1.5 Life expectancy greater than 6 months.
- 3.1.6 Patients capable of childbearing must agree to use adequate contraception.
- 3.1.7 Ability to complete questionnaire(s) by themselves or with assistance.
- 3.1.8 Ability to provide written informed consent.
- 3.1.9 Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).

#### 3.2 Exclusion Criteria

- 3.2.1 Previous radiation therapy to the site of the sarcoma or area surrounding it such that it would be encompassed by the radiation field needed to treat the current sarcoma. In other words, treatment on this trial would require re-irradiation of tissues.
- 3.2.2 Patients with nodal or distant metastases.
- 3.2.3 Rhabdomyosarcoma, soft tissue osteosarcoma, soft tissue Ewing sarcoma, and benign histologies.
- 3.2.4 Any of the following:
  - Pregnant women
  - Nursing women
  - Men or women of childbearing potential who are unwilling to employ adequate contraception

## 4.0 Test Schedule

| | Pre-treatment/ | Нуро- | Post-RT | Pre- | Post- | Years 1 & 2 | Years 3-5 |
|---|---|---|---|---|---|---|---|
| | Baseline | fractionated | Assessment | Operative | Operative | Post-Surgery | Post-Surgery |
| | | RT | | Assessment | Assessment | Assessment | Assessment |
| | | | | | | | Annually Post- |
| | ≤30 days | 42.75 Gy in 15 | (+/- 5 days) | Within 2 | 4-8 weeks | Post- | Surgery <sup>7,8,9</sup> |
| | prior to | fractions | ( ' | weeks of | Post-Surgery6,9 | Surgery <sup>7,8,9</sup> (+/- | (+/- 8 weeks) |
| | registration | J. 272 272 | | surgery <sup>9</sup> | 1 000 | 8 weeks) | ( ' |
| | | | | Su. 80. y | | ĺ | |
| History, physical | | | | | | | |
| exam <sup>7</sup> , ECOG | X | | X | X | | X | X |
| status | 11 | | 11 | 71 | | 11 | 11 |
| Pathology review <sup>1</sup> | X | | | | X | | |
| Primary site MRI <sup>2</sup> , | | | | X | | | |
| 5 | X | | | 11 | | X | X |
| PET/CT or CT | X | | | X | | X | X |
| Chest <sup>5,</sup> | | | | | | Λ | Λ |
| Pregnancy test <sup>3</sup> | X | | | | | | |
| AE Acute | | | | | | | |
| Assessment (See | X | | X | X | | | |
| section 10.0) | | | | | | | |
| Hypofractionated | | X | | | | | |
| RT | | Λ | | | | | |
| CTCAE v5.0 | | | | | | | |
| Solicited Late | X | | | | X | X | X |
| Toxicity | Λ | | | | Λ | Λ | Λ |
| Assessment (See | | | | | | | |
| section 10.0) | | | | | | | |
| Wound | | | | | | | |
| Complication | | | | | | | |
| Assessment | | | | | X | X | |
| (Appendix | | | | | | | |
| VI/Section 11.0) | | | | | | | |
| Regional Alopecia | | | | | | | |
| Assessment | X | | X | X | | | |
| (Appendix V) | | | | | | | |
| Joint Stiffness | | - | | X | | | |
| Assessment | X | | X | | | X | X |
| (Appendix IV) | | | | | | | |
| PROMISE-10 <sup>a</sup> | X | | | X | | X <sup>4</sup> | |
| TESS <sup>b</sup> | X | | | X | | $X^4$ | |

- 1. Pathology review includes histopathologic diagnosis of soft tissue sarcoma and grade, where applicable.
- 2. CT is acceptable if MRI is not advisable.
- 3. For women of childbearing potential only. Must be done ≤7 days prior to beginning radiation treatment. Tubal ligation and IUD in place are exceptions.
- 4. Obtained at 12, 18, and 24 months.
- 5. Within 60 days of enrollment
- 6. Follow Up timepoints may be evaluated outside the anticipated window as deemed appropriate by Stand of Care Radiation Oncology and Orthopedic Surgery follow up schedule
  - a. Patient-Reported Outcomes Measurement Information System
  - b. Toronto Extremity Salvage Score
- 7. Assessments may be completed by NP/PA in person or by virtual and/or phone visit if patient is unable to return to study site.
- 8. Per physician discretion
- 9. If patient develops any type of disease progression or is unwilling to return to the institution, patients will move to yearly survival follow up. No additional assessments will need to be done.

## 5.0 Grouping Factors

5.1 Anatomical Sites of Tumor: Proximal lower extremity (includes knee) versus rest.

Note: As of July 19, 2023, there are no restrictions on number of patients enrolled per anatomical sites of tumor.

## 6.0 Registration Procedures

Patients will be registered by completing the registration through PTrax, and eligibility case report forms (CRFs) stored in MedidataRave.

- 6.1 Prior to patient enrollment, the investigator should ensure that all of the following requirements are met:
  - 6.1.1 The patient meets all inclusion criteria and exclusion criteria apply.
  - 6.1.2 The patient and investigator have signed and dated all applicable consent forms.
  - 6.1.3 All baseline assessments and examinations have been performed.
  - 6.1.4 All registration CRFs have been completed, signed, and dated.
  - 6.1.5 Protocol treatment must begin within 2 weeks of registration.

#### 7.0 Protocol Treatment

## 7.1 Radiation Therapy

All patients enrolled on this trial will receive radiation therapy as detailed below.

#### 7.1.1 Simulation

## 7.1.1.1 Patient Positioning and Immobilization

The patient may be treated in any appropriate, stable position. No specific immobilization is mandated. However, reproducible setup is critical and the use of standard immobilization devices for the extremity and/or truck is strongly encouraged.

Bolus should not be used unless:

- a. The tumor involves cutaneous structures,
- b. The tumor is very superficial such that adequate target dose (<90% prescription dose to the planning target volume (PTV)) cannot be delivered without it,
- c. Or, the surgeon indicates the biopsy scar and/or skin will not be resected.

#### 7.1.1.2 Image Acquisition

Computed tomography (CT) imaging obtained during simulation will be the primary imaging modality for target delineation and

treatment planning. CT simulation imaging will be obtained per institutional policies and procedures.

Diagnostic or treatment position Magnetic Resonance Imaging (MRI) may be used to aid with target delineation and treatment planning at the discretion of the treating radiation oncologist. Similarly, use of intravenous contrast, breath hold techniques, and acquisition of 4D imaging sets are at the discretion of the treating radiation oncologist.

## 7.1.2 Target Volume Definitions

Treatment planning will be based on the following definitions.

#### 7.1.2.1 GTV

Gross tumor volume (GTV) is the volume of all known disease based on CT simulation imaging and physical exam. If MRI is used for target delineation, GTV is best delineated on T1 contrast sequences.

If there has been prior surgical violation of the sarcoma (for example, a non-oncologic partial or positive-margin excision), the GTV may be extended to include the initial region of gross tumor as well as any disturbed tissues. In most cases, an open biopsy scar should not be included in the GTV as standard of care is for the incision to be resected. In the unusual situation where an open biopsy scar will not be resected, this should be confirmed with the surgeon and included in the GTV.

### 7.1.2.2 CTV

Clinical target volume (CTV) includes the GTV and sites of potential occult tumor involvement. A 2.0-4.0 cm longitudinal and 1.0-1.5 cm radial expansion from GTV will be used to generate the CTV. The expansions should follow natural planes of spread for sarcomas, while respecting intact bone and compartment boundaries. If MRI is used for target delineation, the CTV should also include physician-determined suspicious peri-tumoral edema seen on T2 sequence images. In patients who received neoadjuvant chemotherapy and experienced a reduction in tumor volume with chemotherapy, the pre-chemotherapy extent of the tumor in soft tissues should be included in the CTV.

#### 7.1.2.3 PTV

A geometric margin of 5-10 mm will be used to create PTV. Daily image guidance is required.

## 7.1.2.4 Proton Therapy

- 7.1.2.4.1 GTV is the same for protons and photons
- 7.1.2.4.2 CTV is the same for protons and photons
- 7.1.2.4.3 PTV is not the same as photons due to differences in beam penetration with movement and set up uncertainty. PTV varies with each individual field and requires additional adjustments based on set up error for the involved body site. In general, adjustment margins are usually 2-7 mm and will follow institutional policies and procedures.

## 7.1.3 Organs at Risk Contouring Definitions

Only organs at risk relevant to the treatment field within 2 cm superior and inferior to the PTV edge should be contoured.

- 7.1.3.1 Bone avoid (only applicable for extremity tumors)

  The bone immediately adjacent to the gross tumor is contoured as bone avoid. The bone avoid structure will extend 2 cm superior and inferior to the PTV edge.
- 7.1.3.2 Soft tissue avoid (only applicable for extremity tumors)

  The soft tissue surrounding the PTV and extending 2 cm superior and inferior to the PTV edge is defined as soft tissue avoid. To create the soft tissue avoid structure, an intermediate structure is first created defined as PTV + a 2.0 cm geometric expansion.

  Then, the body only contour is subtracted from the PTV+2.0 cm intermediate structure and limited to 2 cm superior and inferior to the PTV edge. This final soft tissue avoid structure is cropped out of bone avoid and volumes <1cm³ are erased (Figure 1).

Figure 1. Example of the soft tissue avoid structure in axial plane. PTV is in magenta, soft tissue avoid is in light green, and bone avoid is in orange.



## 7.1.4 Radiation Therapy Planning

#### 7.1.4.1 Dose definition

Photon dose will be specified in centigray (cGy). For proton therapy, the absorbed dose is specified in centigray equivalents (CGE), which is the same as ICRU 78  $D_{RBE}$  using a standard RBE of 1.10 with respect to water.

#### 7.1.4.2 Target Dose

The radiation dose prescribed to the PTV will be 4275 cGy in 15 daily fractions over 3 weeks. Treatment will be delivered once daily, except on weekends and holidays. Twice daily (BID) treatments are not allowed.

#### 7.1.4.3 Treatment Planning

The treatment technique and modality are at the discretion of the treating radiation oncologist. The patient may be treated using conventional 3D radiotherapy (3DCRT); Intensity Modulated Radiotherapy (IMRT), rotational IMRT techniques such as Volumetric Arc Radiation Therapy (VMAT), or proton therapy (3D or Intensity Modulated Proton Therapy (IMPT)).

The dose will be prescribed to the treatment isocenter, which serves as the ICRU reference point. Appropriate beam modality and energy should be selected for the size and depth of the tumor, tissue, and site to be treated. Every attempt should be made to use techniques (i.e., 3DRT, IMRT, VMAT, etc.) and modalities (i.e.,

electrons, photons, protons) which avoid unnecessary irradiation of critical normal tissues.

7.1.4.4 Target Dose Requirements and Uniformity
Table 1.0 lists dose volume histogram (DVH) requirements for
CTV and PTV. If DVH requirements cannot be met, an
explanation must be submitted to the study co-chairs (S. K.
Ahmed, M.D. or I.A. Petersen, M.D.).

Table 1.0 – DVH requirements for CTV and PTV

| Structure | DVH<br>Endpoint | Requirement | Priority | DVH<br>Endpoint | Requirement | Priority |
|---|---|---|---|---|---|---|
| CTV_4275 | D95%[%] | ≥ 100% | 2 | D95%[%] | ≥ 95% | 1 |
| | | | | CV95%[cc] | <0.5cc | 1 |
| | V110% | | Report | | | |
| PTV_4275 | D95%[%] | ≥ 99% | 2 | D95%[%] | ≥ 95% | 1 |
| | | | | CV95%[cc] | <0.5 cc | 1 |
| | V110% | | Report | | | |

## 7.1.4.4.1 Minor Deviation Definition

a) PTV\_4275 D95% <95% but  $\ge$  90%

AND / OR

b) >20% but ≤ 25% of PTV\_4275 receives ≥110% of prescription dose

## 7.1.4.4.2 Major Deviation Definition

a) PTV 4275 D95% <90%

AND / OR

b) >25% of PTV\_4275 receives ≥110% of prescription dose

AND/OR

c) Dose to the priority 1 organs at risk is more than the recommended limit (Table 2.0)

## 7.1.4.5 Organs at Risk Dose Constraints

Normal tissue dose constraints are listed in Table 2.0. Every effort should be made to avoid treating the full circumference of any extremity. There is no special requirement for skin dose limit. However, full prescription dose to skin over areas commonly traumatized (e.g., elbow, knee, shin) should be avoided unless in the PTV.

While every effort should be made to deliver prescription doses to the PTV as specified while adhering to normal tissue constraints, it is recognized that certain anatomical factors may prevent this. As such, if normal tissue constraints are unachievable, the patient will be taken off the trial and treated with standard pre-operative RT to 50 Gy in 25 fractions meeting standardly accepted constraints for that fractionation schedule.

Table 2.0 –Organs at Risk Dose Constraints

| Organ at Risk | Dose Constraints | Priority |
|---|---|---|
| Bone avoid | Mean < 32 Gy | 1 |
| | V35Gy < 64% | 1 |
| | V35Gy < 40% | 2 |
| Soft tissue avoid | Mean < 26 Gy | 2 |
| | V18Gy <50% | 1 |
| Joint (only major joints:<br>hip/knee/shoulder) | V42.56Gy <50% | 2 |
| Anus | Max | Report |
| | V42.75Gy (%) | Report |
| | V40.6Gy (%) | Report |
| Genitalia | Max | Report |
| | Mean <26 Gy | 1 |

| Testis (if fertility preservation | V1Gy ≤ 60% | 1 |
|---|---|---|
| desired) | V1Gy ≤ 50% | 2 |
| Ovaries (if fertility | V4.8Gy ≤ 60% | 1 |
| preservation desired) | V1Gy ≤ 50% | 2 |
| Lungs | V18Gy≤ 20% | 1 |
| Brachial plexus | Max < 48 Gy | 1 |
| Heart | Mean < 10 Gy | 1 |
| Esophagus | Mean <26 Gy | 1 |
| Liver | Mean <26 Gy | 1 |
| Stomach | Max ≤38 Gy | 1 |
| Small Bowel | Max ≤ 45 Gy; if in PTV | 21 |
| | V42.75Gy <20 cc | 2 |
| | V26.5Gy <100 cc | 1 |
| | V39Gy <60 cc | |
| Large Bowel | Max < 45 Gy; if in PTV | 2Report |
| | V42.75Gy (%) | Report |
| | V40.6Gy (%) | 2 |
| | V42.75Gy (cc) <50 cc | |
| Kidney | V11.8 Gy < 10% for total kidney volume | 1 |
| | V11.8Gy <33% for each kidney | 2 |
| | V5Gy for each kidney | Report |
| Spinal Cord | Max | Report |

| | V39Gy <0.1% | 2 |
|---------|---------------|--------|
| Bladder | Max | Report |
| | V42.75Gy <50% | 2 |
| | V30Gy <60% | 2 |

## 7.1.5 Radiation Therapy Delivery

Radiation therapy will be delivered using a linear accelerator or proton gantry. Patients will be set up according to the instructions from CT simulation and treatment planning. Image guidance procedures will be determined at the discretion of the treating radiation oncologist.

## 7.1.6 Treatment Delays

There will be no planned rests or breaks from treatment. Once radiation therapy has been initiated, treatment will not be interrupted except for severe illness or unplanned emergencies. The reason for any interruptions greater than three days should be recorded and submitted to the study Chair (S.K. Ahmed, M.D.). When treatment interruptions or delays occur, the total number of fractions or cumulative dose should not be modified.

## 7.1.7 Special Considerations

#### 7.1.7.1 Tumor motion

Acquisition of 4D imaging sets, use of breath hold techniques, or treatment delivery via phase gating for tumors with internal motion are at the discretion of the treating radiation oncologist. In these cases, an internal target volume (ITV) will be delineated per standard institutional policies and procedures.

#### 7.1.7.2 Nodal Radiation

For tumors with no evidence of nodal involvement, the draining regional lymph nodes should not be irradiated. Tumors with nodal involvement are excluded on this trial.

#### 7.1.8 Quality Assurance

All target volumes and final treatment plans must be submitted for review and approval by a study co-chair (S. K. Ahmed, M.D. or I.A. Petersen, M.D.).

## 7.1.9 Intraoperative and Postoperative Radiation Therapy

Use of intraoperative and postoperative radiation therapy is discouraged. If intraoperative or postoperative radiation therapy is deemed to be of benefit for a high-risk case, contact a study co-chair (S. K. Ahmed, M.D. or I.A. Petersen, M.D.).

## 7.2 Surgery

Patients will undergo oncologic resection ideally 3-4 weeks after completion of preoperative radiation therapy per institutional standards. If surgery is not feasible during this ideal period, it must be performed within 6 weeks ( $\pm$  1 week) of completing preoperative radiation therapy. Acute wound complications will be recorded as detailed in section 11.1.

20

## 7.3 Chemotherapy

The use of chemotherapy will be at the discretion of the multidisciplinary team and medical oncology consultant involved in the case. Chemotherapy will not be used concurrently with radiation therapy on this study. In cases where chemotherapy is used either neo-adjuvantly or adjuvantly, the agents used and number of cycles/doses of chemotherapy will be documented.

## 7.4 Patient reported questionnaires

All patients will complete Patient-Reported Outcomes Measurement Information System (PROMIS) and Toronto Extremity Salvage Score (TESS) questionnaires at baseline, post-radiotherapy, and post-surgery time-points as detailed in section 4.0.

## 8.0 Dosage Modifications Based on Adverse Events

N/A

## 9.0 Ancillary Treatment/Supportive Care

## 9.1 Permitted Supportive Therapy

All supportive therapies for optimal medical care are allowed during the study period at the discretion of the provider within the parameters of the protocol. Examples include skin care, physical therapy and rehabilitation, occupational therapy, antiemetics, anti-diarrheals, prophylaxis for constipation, anti-inflammatories, antipyretics, intravenous fluids, and appetite enhancers.

## 9.2 Non-permitted Supportive Therapy

No investigational agents are permitted.

#### 10.0 Adverse Event (AE) Monitoring and Reporting

#### 10.1 Definitions

<u>Adverse Event</u>- An untoward or undesirable experience associated with the use of a medical product (i.e. drug, device, biologic) in a patient or research subject.

Serious Adverse Event – Any grade 4 or 5 adverse event as defined by CTCAE v5.0. Adverse events are classified as serious or non-serious. Serious problems/events can be well defined and include in general:

- Death
- Life threatening adverse experience where emergent lifesaving treatment is necessary.

<u>Unanticipated Problems Involving Risks to Subjects or Others (UPIRTSO)</u>- Any unanticipated problem or adverse event that meets the following three criteria:

Serious: Serious problems or events that results in significant harm, (which may be physical, psychological, financial, social, economic, or legal) or increased risk for the subject or others (including individuals who are not research subjects). These include: (1) death; (2) life threatening adverse experience; (3) hospitalization - inpatient, new, or prolonged; (4) disability/incapacity - persistent or significant; (5) birth defect/anomaly; (6) breach of confidentiality and (7) other problems, events, or new information (i.e. publications, DSMB reports, interim findings, product labeling change) that in the opinion of the local investigator may adversely affect the rights, safety, or welfare of the subjects or others, or substantially compromise the research data,

#### AND

<u>Unanticipated</u>: (i.e. unexpected) problems or events are those that are not already described as potential risks in the protocol, consent document, not listed in the Investigator's Brochure, or not part of an underlying disease. A problem or event is "unanticipated" when it was unforeseeable at the time of its occurrence. A problem or event is "unanticipated" when it occurs at an increased frequency or at an increased severity than expected,

#### **AND**

<u>Related</u>: A problem or event is "related" if it is possibly related to the research procedures.

<u>Preexisting Condition</u>- A preexisting condition is one that is present at the start of the study. A preexisting condition should be recorded as an adverse event if the frequency, intensity, or the character of the condition worsens during the study period. At screening, any clinically significant abnormality should be recorded as a preexisting condition. At the end of the study, any new clinically significant findings/abnormalities that meet the definition of an adverse event must also be recorded and documented as an adverse event.

## 10.2 Recording Adverse Events

CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events

(CTCAE) version 5.0 will be utilized for AE reporting unless as otherwise stated in the table below.

All appropriate treatment areas should have access to a copy of the CTCAE version 5.0. A copy of the CTCAE version 5.0 can be downloaded from the CTEP web site:

(http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm)

10.2.1 Adverse event monitoring and reporting is a routine part of every clinical trial. First, identify and grade the severity of the event using the CTCAE version 5.0. Next, determine whether the event is expected or unexpected and if the adverse event is related to the medical treatment or procedure. With this information, determine whether the event must be reported as an expedited report (see Section 10.3).

#### 10.2.2 Assessment of Attribution

Only G4 or G5 adverse events will require an attribution. Any change in the grade of an adverse event within the list of monitored AEs will be recorded and considered to be related to treatment. Any new adverse not listed occurring within the radiated area or in close proximity will be graded and attribution defined by the study PI. Events determined to be possibly, probably or definitely attributed to a medical treatment suggest there is evidence to indicate a causal relationship between the treatment and the adverse event.

## 10.3 Reporting of Serious Adverse Events and Unanticipated Problems

When an adverse event has been identified, the study team will take appropriated action necessary to protect the study participant and then complete the Study Adverse Event Worksheet and log. The sponsor-investigator will evaluate the event and determine the necessary follow-up and reporting required.

a. Serious Adverse Events will be reported as part of regular adverse event reporting mechanisms via the data capture system and logged for review reporting.

## 10.3.1 Investigator Reporting: Notifying the Mayo IRB

The IRB requirements reflect the guidance documents released by the Office of Human Research Protections (OHRP), and the Food and Drug Administration (FDA) in early 2007 and are respectively entitled "Guidance on Reviewing and Reporting Unanticipated Problems Involving Risks to Subjects or Others and Adverse Events" and "Guidance for Clinical Investigators, Sponsors, and IRBs: Adverse Event Reporting – Improving Human Subject Protection."

10.3.1.1 According to Mayo IRB Policy any serious adverse event (SAE) which the Principal Investigator has determined to be a UPIRTSO must be reported to the Mayo IRB as soon

as possible but no later than 5 working days after the investigator first learns of the problem/event.

10.3.1.2 Non-UPIRTSO – the investigator reports problems or events that do NOT meet criteria of an UPIRTSO in summary format at the time of the next continuing review. The investigator monitors the severity and frequency of subsequent non-UPIRTSOs.

Consider the following information to collect when developing any forms for documentation of adverse events.

## **Example**

Information collected on the adverse event worksheet (and entered in the research database):

- Subject's name:
- Medical record number:
- Disease/histology (if applicable):
- The date the adverse event occurred:
- Description of the adverse event:
- Relationship of the adverse event to the research (drug, procedure, or intervention):
- If the adverse event was expected:
- The severity of the adverse event: (use a table to define severity scale 1-5)
- If any intervention was necessary:
- Resolution: (was the incident resolved spontaneously, or after discontinuing treatment)
- Date of Resolution:

The investigator will review all adverse event reports to determine if specific reports need to be made to the IRB and FDA. The investigator will sign and date the adverse event report when it is reviewed. For this protocol, only directly related SAEs/UPIRTSOs will be reported to the IRB.

10.4 Solicited toxicities to be graded at each evaluation and pretreatment symptoms/conditions to be evaluated based on the schedule of events using the CTCAE v5.0 grading unless otherwise stated in the table below. This regimen has established safety, based on this article <a href="https://www.thelancet.com/journals/lanonc/article/PIIS1470-2045(22)00638-6/fulltext">https://www.thelancet.com/journals/lanonc/article/PIIS1470-2045(22)00638-6/fulltext</a> so the focus is on solicited toxicities and not any adverse event after radiation therapy is completed.

| ACUTE TOXICITIES – Upper Proximal Extremity | | | |
|---|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event /<br>Symptoms | Baseline | During RT & Preoperative Assessment |

| General disorders and administration site conditions | Fatigue | X | X |
|---|---|---|---|
| Skin and subcutaneous tissue | Dermatitis<br>Radiation | X | X |
| disorders | Hyperpigmentation | X | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain | X | X |

| LATE TOXICITIES – Upper Proximal Extremity | | |
|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event / Symptoms | Post-Surgery & Follow Up |
| Skin and subcutaneous tissue disorders | Hyperpigmentation <sup>1</sup> | X |
| Vascular | Lymphedema <sup>2</sup> | X |
| General disorders and administration site conditions | Localized edema <sup>1</sup> | X |
| Musculoskeletal and connective tissue | Fibrosis deep connective tissue <sup>1</sup> | X |
| disorders | Joint range of motion decreased <sup>2</sup> | X |
| | Osteonecrosis <sup>1</sup> | X |

| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain <sup>1</sup> | X |
|---|---|---|
| Injury, poisoning and procedural complications | Fracture <sup>1</sup> | X |
| Gastrointestinal Disorders <sup>1</sup> | Esophageal fistula | X |
| Respiratory, thoracic and mediastinal disorders | Pneumonitis <sup>1</sup> | X |

<sup>&</sup>lt;sup>1</sup> Specific to radiation / surgery treatment area
<sup>2</sup> Specific to ipsilateral extremity / region

| <b>ACUTE TOXICITIES – Upper Distal Extremity (includes elbow)</b> | | | |
|---|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event /<br>Symptoms | Baseline | During RT & Preoperative Assessment |
| General disorders<br>and administration<br>site conditions | Fatigue | X | X |
| Skin and subcutaneous tissue | Dermatitis<br>Radiation | X | X |
| disorders | Hyperpigmentation | X | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain | X | X |

| LATE TOXICITIES – Upper Distal Extremity (includes elbow) | | |
|---|---|---|
| CTCAE System/Organ/Class (SOC) | Adverse Event / Symptoms | Post-Surgery & Follow Up |
| Skin and subcutaneous tissue disorders | Hyperpigmentation <sup>1</sup> | X |
| Vascular | Lymphedema <sup>2</sup> | X |
| General disorders and administration site conditions | Localized edema <sup>1</sup> | X |
| Musculoskeletal and connective tissue | Fibrosis deep connective tissue <sup>1</sup> | X |
| disorders | Joint range of motion decreased <sup>2</sup> | X |
| | Osteonecrosis <sup>1</sup> | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain <sup>1</sup> | X |
| Injury, poisoning and procedural complications | Fracture <sup>1</sup> | X |

| ACUTE TOXICITIES – Lower Proximal Extremity (includes knee) | | | |
|---|---|---|---|
| CTCAE System/Organ/Class (SOC) | Adverse Event /<br>Symptoms | Baseline | During RT & Preoperative<br>Assessment |
| General disorders<br>and administration<br>site conditions | Fatigue | X | X |

| Skin and subcutaneous tissue disorders | Dermatitis<br>Radiation | X | X |
|---|---|---|---|
| | Hyperpigmentation | X | X |
| | Diarrhea | X | X |
| Gastrointestinal disorders | Nausea | X | X |
| disorders | Vomiting | X | X |
| Renal and urinary disorders | Dysuria | X | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain | X | X |

| LATE TOXICITIES – Lower Proximal Extremity (includes knee) | | |
|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event /<br>Symptoms | Post-Surgery & Follow Up |
| Skin and subcutaneous tissue disorders | Hyperpigmentation <sup>1</sup> | X |
| Vascular | Lymphedema <sup>2</sup> | X |
| General disorders and administration site conditions | Localized edema <sup>1</sup> | X |
| | Fibrosis deep connective tissue <sup>1</sup> | X |

| Musculoskeletal and connective tissue disorders | Joint range of motion decreased <sup>2</sup> | X |
|---|---|---|
| disorders | Osteonecrosis <sup>1</sup> | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain <sup>1</sup> | X |
| Injury, poisoning and procedural complications | Fracture <sup>1</sup> | X |
| Gastrointestinal Disorders <sup>1</sup> | Anal fistula | X |
| Disorders | Colonic fistula | X |
| | Duodenal fistula | X |
| | Ileal fistula | X |
| | Jejunal fistula | X |
| | Rectal fistula | X |
| | Anal ulcer | X |
| | Colonic ulcer | X |
| | Duodenal ulcer | X |
| | Ileal ulcer | X |
| | Jejunal ulcer | X |
| | Rectal ulcer | X |
| | Small intestine ulcer | X |
| | Anal stenosis | X |
| | Colonic stenosis | X |
| | Duodenal stenosis | X |

| | Ileal stenosis | X |
|------------------------------------------|-----------------------------|---|
| | Jejunal stenosis | X |
| | Rectal stenosis | X |
| | Small intestine stenosis | X |
| | Rectal perforation | X |
| | Small intestine perforation | X |
| | Colonic perforation | X |
| | Duodenal perforation | X |
| | Ileal perforation | X |
| | Jejunal perforation | X |
| | Enterovesical fistula | X |
| Renal and urinary disorders <sup>1</sup> | Urinary fistula | X |
| disorders | Bladder perforation | X |

<sup>&</sup>lt;sup>1</sup> Specific to radiation / surgery treatment area <sup>2</sup> Specific to ipsilateral extremity / region

| A | CUTE TOXICITIES | 5 – Lower Dista | l Extremity |
|---|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event /<br>Symptoms | Baseline | During RT & Preoperative Assessment |

| General disorders and administration site conditions | Fatigue | X | X |
|---|---|---|---|
| Skin and subcutaneous tissue | Dermatitis<br>Radiation | X | X |
| disorders | Hyperpigmentation | X | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain | X | X |

<sup>&</sup>lt;sup>1</sup> Per study definition

| LATE TOXICITIES – Lower Distal Extremity | | |
|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event / Symptoms | Post-Surgery & Follow Up |
| Skin and subcutaneous tissue disorders | Hyperpigmentation <sup>1</sup> | X |
| Vascular | Lymphedema <sup>2</sup> | X |
| General disorders and administration site conditions | Localized edema <sup>1</sup> | X |
| Musculoskeletal and | Fibrosis deep connective tissue <sup>1</sup> | X |
| connective tissue<br>disorders | Joint range of motion decreased <sup>2</sup> | X |
| | Osteonecrosis <sup>1</sup> | X |

| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain <sup>1</sup> | X |
|---|---|---|
| Injury, poisoning and procedural complications | Fracture <sup>1</sup> | X |

<sup>&</sup>lt;sup>1</sup> Specific to radiation / surgery treatment area <sup>2</sup> Specific to ipsilateral extremity / region

| ACUTE TOXICITIES – Superficial Trunk | | | |
|---|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event /<br>Symptoms | Baseline | During RT & Preoperative<br>Assessment |
| General disorders<br>and administration<br>site conditions | Fatigue | X | X |
| Skin and subcutaneous tissue disorders | Dermatitis<br>Radiation | X | X |
| | Hyperpigmentation | X | X |
| Gastrointestinal disorders | Diarrhea | X | X |
| | Nausea | X | X |
| | Vomiting | X | X |
| Renal and urinary disorders | Dysuria | X | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain | X | X |

| LATE TOXICITIES | | |
|---|---|---|
| CTCAE<br>System/Organ/Class<br>(SOC) | Adverse Event / Symptoms | Post-Surgery & Follow Up |
| Skin and subcutaneous tissue disorders | Hyperpigmentation <sup>1</sup> | X |
| General disorders and administration site conditions | Localized edema <sup>1</sup> | X |
| | Lymphedema | X |
| Musculoskeletal and connective tissue disorders | Fibrosis deep connective tissue <sup>1</sup> | X |
| | Joint range of motion decreased <sup>2</sup> | X |
| | Osteonecrosis <sup>1</sup> | X |
| Neoplasm benign,<br>malignant and<br>unspecified | Tumor pain <sup>1</sup> | X |
| Injury, poisoning and procedural complications | Fracture <sup>1</sup> | X |
| Gastrointestinal Disorders <sup>1</sup> | Anal fistula | X |
| | Colonic fistula | X |
| | Duodenal fistula | X |
| | Esophageal fistula | X |
| | Gastric fistula | X |
| | Ileal fistula | X |
| | Jejunal fistula | X |

| Rectal fistula | X |
|-----------------------------|---|
| Anal ulcer | X |
| Colonic ulcer | X |
| Duodenal ulcer | X |
| Gastric ulcer | X |
| Ileal ulcer | X |
| Jejunal ulcer | X |
| Rectal ulcer | X |
| Small intestine ulcer | X |
| Anal stenosis | X |
| Colonic stenosis | X |
| Duodenal stenosis | X |
| Gastric stenosis | X |
| Ileal stenosis | X |
| Jejunal stenosis | X |
| Rectal stenosis | X |
| Small intestine stenosis | X |
| Rectal perforation | X |
| Small intestine perforation | X |
| Colonic perforation | X |
| Duodenal perforation | X |
| Gastric perforation | X |
| Ileal perforation | X |

| | Jejunal perforation | X |
|---|---|---|
| | Enterovesical fistula | X |
| Renal and urinary disorders <sup>1</sup> | Urinary fistula | X |
| disorders | Bladder perforation | X |
| Respiratory, thoracic and mediastinal disorders | Pneumonitis <sup>1</sup> | X |

<sup>&</sup>lt;sup>1</sup> Specific to radiation / surgery treatment area

- 10.5 Submit via appropriate *reporting mechanisms* the following AEs experienced by a patient through the course of Radiation Therapy and not specified in Section 10.4:
  - 10.5.1 Grade 3, 4, and 5 AEs regardless of attribution to the study treatment or procedure.
  - 10.5.2 Grade 5 AEs (Death)
    - 10.5.2.1 Any death within 30 days of the patient's last study treatment or procedure regardless of attribution to the study treatment or procedure
    - 10.522 Any death more than 30 days after the patients last study treatment or procedure that is felt to be at least possibly treatment related must also be submitted as a Grade 5 AE, with a CTCAE type and attribution assigned.

## 10.6 Monitoring and Auditing

The investigator will permit study-related monitoring, audits, and inspections by the IRB, the sponsor, and government regulatory agencies, of all study related documents (e.g. source documents, regulatory documents, data collection instruments, study data etc.). The investigator will ensure the capability for inspections of applicable study-related facilities (e.g. pharmacy, diagnostic laboratory, etc.). Participation as an investigator in this study implies acceptance of potential inspection by government regulatory authorities and applicable compliance offices.

#### 10.6.1 Medical Monitoring

<sup>&</sup>lt;sup>2</sup> Specific to ipsilateral extremity / region

It is the responsibility of the Principal Investigator to oversee the safety of the study at his/her site. This safety monitoring will include careful assessment and appropriate reporting of adverse events as noted above, as well as the construction and implementation of a site data and safety-monitoring plan (see section 10.5 "Monitoring and Auditing"). Medical monitoring will include a regular assessment of the number and type of serious adverse events. Any serious adverse events will be followed up by the sentinel event reporting procedure.

## 10.6.2 Internal Data and Safety Monitoring Board

The trial will be reviewed by the Cancer Center Auditing area on a biannual or yearly basis dependent on random study selection to assess accrual, adverse events, and any endpoint problems. Any safety issues requiring protocol changes will be communicated through protocol amendments.

#### 11.0 Treatment Evaluation/Measurement of Effect

- 11.1 Development of a surgical wound complication: Secondary unplanned operation under general or regional anesthesia for wound repair (e.g., debridement, operative drainage, or secondary wound closure including rotationplasty, free flaps or skin grafts); or wound management without secondary operation including invasive procedures (e.g., aspiration of seroma or readmission for wound care such as intravenous antibiotics or persistent deep packing for 120 days or longer).
- 11.2 Local recurrence free survival: Any radiographic or pathologic evidence of recurrent disease inside the CTV and/or beyond the CTV to within a 3 cm distance from the edge of the CTV. Ideally assessed by radiographic imaging in comparison to the treatment fields in order to determine site of recurrence.

#### 12.0 Descriptive Factors

- 12.1 ECOG Performance Status: 0 versus 1 versus 2 versus 3.
- 12.2 Sex: Male versus female.
- 12.3 Age: 18-30 versus 31-50 versus 51-70 versus  $\geq 70$ .
- 12.4 Tumor Size: <5 cm versus 5-10 cm versus 11-15 cm versus >15 cm.
- 12.5 Anatomic location: Proximal upper extremity versus distal upper extremity (including elbow) versus proximal lower extremity (including knee) versus distal lower extremity versus superficial trunk.
- 12.6 Lesion presentation: de novo (biopsy only) versus status post inadvertent excision.
- 12.7 Histology: Undifferentiated pleomorphic sarcoma versus liposarcoma versus leiomyosarcoma versus myxofibrosarcoma versus other histology.
- 12.8 Tumor depth: Superficial and deep to fascia versus deep to fascia versus superficial to fascia.
- 12.9 Radiation Treatment Modality: 3D conformal versus IMRT versus proton therapy.
- 12.10 Neoadjuvant chemotherapy: Yes versus no.
- 12.11 Margin status: R0 vs R1 vs R2.
- 12.12 Surgical closure: Primary closure versus skin graft versus flap.

#### 13.0 Treatment / Follow-up Decision at Evaluation of Patient

As per standard of care, throughout the study, investigators can prescribe any medications/treatments that have been deemed necessary for the well-being and over all treatment of the patient.

- 13.1 A patient is deemed ineligible if after registration, it is determined that at the time of registration, the patient did not satisfy each and every eligibility criteria for study entry. The patient will go off study.
  - If the patient received MR for radiotherapy planning, all data up until the point of confirmation of ineligibility must be submitted.
  - If the patient never received radiation therapy, on-study material must be submitted. No additional follow up is necessary.
- 13.2 Those patients who will not receive any radiation treatment or who will receive radiation treatment elsewhere will go off study.
- 13.3 Inevaluable Patients

If a patient fails to complete radiation therapy for reasons other than toxicity, the patient will be regarded as inevaluable and will be replaced.

13.4 Patients with a Major Deviation

AND / OR

A patient is deemed a major violation if:

a) PTV\_4275 D95% <90%

MC1973

b) >25% of PTV\_4275 receives  $\geq$ 110% of prescription dose AND / OR

37

c) Dose to the organs at risk is more than the recommended limit (Table 2.0) These patients will be flagged but included in the primary endpoint analysis. Separate sensitivity analysis will also be performed between the patients with major violation vs no major violation on major wound complication rate.

#### 14.0 Body Fluid Biospecimens

N/A

#### 15.0 Drug Information

N/A

#### 16.0 Statistical Considerations and Methodology

#### 16.1 Overview

This phase II single arm study will utilize a non-inferiority design approach to assess the rate of major wound complications associated with hypofractionated preoperative radiation therapy of 42.75 Gy in 15 fractions for localized, resectable soft tissue sarcoma of the extremity and superficial trunk compared to conventional fractionation of 50 Gy in 25 fractions.

## 16.1.1 Primary Endpoint

The primary endpoint of this trial is the proportion of patients who experience major wound complications within 120 days of surgical resection of soft tissue sarcoma of the extremity and superficial trunk following preoperative radiation therapy of 42.75 Gy in 15 fractions. Major wound complication is defined as secondary unplanned operation under general or regional anesthesia for wound repair (e.g., debridement, operative drainage, or secondary wound closure including rotation plasty, free flaps or skin grafts); or wound management without secondary operation including invasive procedures (e.g., aspiration of seroma or readmission for wound care such as intravenous antibiotics or persistent deep packing for 120 days or longer). All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for the primary endpoint.

#### 16.2 Statistical Design

The non-inferiority one-sample test was utilized from PASS software for this design (Non-Inferiority of One Proportion using the Z-Test with S(P0) in PASS 16.0.4). A sample size of 108 evaluable patients achieves 80% power (1-sided significance level of 10%) to detect a non-inferiority margin of 10%, assuming that any major wound complication rate of 45% or above is inferior as compared to the current standard of care complication rate of 35%. We hypothesize that the proposed hypofractionated preoperative radiation therapy of 42.75 Gy in 15 fractions is not inferior to the conventional fractionation of 50 Gy in 25 fractions

by showing the complication rate is < 45% for the proposed treatment (non-inferiority margin of 10%).

#### 16.2.1 Decision Rule

After the first 108 eligible patients have completed 120 days post-treatment, we'll do the final analysis of the data, and if the Z-test is significant at the 10% significance level, we'll conclude that hypofractionated preoperative radiation therapy of 42.75 Gy in 15 fractions is not inferior to conventional fractionation of 50 Gy in 25 fractions and can be tested further in larger studies.

#### 16.2.2 Sample Size

This study is expected to need to accrue 108 evaluable patients unless the study is closed early for excessive toxicity. We anticipate approximately 10% lost to follow-up due to 120 day endpoint, therefore we anticipate accruing an additional 12 patients to account for ineligibility, cancellation, or other reasons, making the overall sample size of 120 patients.

#### 16.2.3 Accrual Rate and Study Duration

The expected accrual rate is about 4 patients per month. With this accrual rate, we expect to finish accrual within about 30 months of study activation, assuming we accrue 120 total patients. The final analysis can begin as soon as the last patient has been observed for 4 months post treatment, or at approximately 3 years after the study opens to accrual.

#### 16.2.4 Power and Significance Level

Assuming that the number of major wound complications is binomially distributed, the significance level is 0.1 i.e. there is 10% chance of finding hypofractionated preoperative radiation therapy to be effective when it truly is not. The probability of declaring that the proposed radiation therapy warrants further studies (i.e., statistical power) is 80.01%, if the true acute wound complication is <45%.

#### 16.2.5 Other Considerations

Adverse events, quality/duration of response, and patterns of treatment failure observed in this study, as well as scientific discoveries or changes in standard care will be taken into account in any decision to terminate the study.

#### 16.3 Analysis Plan

The analysis for this trial will commence at planned time points (see 16.2.3) and at the time the patients have become evaluable for the primary endpoint. The Statistician and Study Chair will make the decision, in accord with CCS Standard Operating Procedures, availability of data for secondary endpoints (e.g., disease free survival, overall survival), and the level of data maturity. It is anticipated that the earliest date in which the results will be made available via manuscript, abstract, or presentation format is when last patient has been followed for at least 6 months.

Note: Both primary and secondary outcomes will be compared between anatomical sites (proximal lower limb (includes knee) vs rest). The comparison between groups will be exploratory in nature.

#### 16.3.1 Primary Outcome Analysis

- 16.3.1.1 Definition: The primary endpoint of this trial is the proportion of patients who experience major wound complications within 120 days of surgical resection of soft tissue sarcoma following preoperative radiation therapy. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for the major wound complication rate.
- 16.3.1.2 Estimation: The proportion of major wound complications will be estimated by the number of patients who experience the major wound complications within 120 days following surgery divided by the total number of evaluable patients. 95% confidence intervals using normal approximation to binomial wound complication proportion will be calculated.
- 16.3.1.3 Over Accrual: If more than the target number of patients are accrued, the additional patients will not be used to evaluate the stopping rule or used in any decision making process; however, they will be included in final endpoint estimates and confidence intervals.

#### 16.3.2 Secondary Outcome Analysis

16.3.2.1 Local failure is defined any radiographic or pathologic evidence of recurrent disease inside the CTV and/ or to within 3 cm from the edge of the CTV. In the absence of censored patients prior to 5 years, local failure rate at 5 years (LFR5) will be equal to the binomial proportion. LFR5 will be evaluated by the number of patients free of local failure/recurrence at 5 year divided by the total number of evaluable patients. Exact binomial 95%

- confidence interval for the point estimate will be provided. In the case of censoring prior to 5 years, LFR5 will be estimated using the Kaplan-Meier method.
- 16.3.2.2 Disease-Free Survival is defined as the time from registration date to the earliest date of documentation of either, local recurrence, regional recurrence, distant recurrence, or death due to any cause, censoring patients who are alive and local recurrence free at the date of last know clinical assessment. The distribution of disease-free survival will be estimated using method of Kaplan-Meier.
- 16.3.2.3 Overall Survival is defined as the time from registration date to death due to any cause, censoring patients alive at the date of last contact. The distribution of overall survival will be estimated using method of Kaplan-Meier.
- 16.3.2.4 Late toxicity is defined as toxicity occurs any time between 3 months and 24 months after completion of hypofractionated preoperative radiation therapy. The rate of ≥ grade 2 late toxicities will be estimated by the number of patients with a ≥ grade 2 late toxicity divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true rate of ≥ grade 2 toxicity events will be calculated.
- 16.3.2.5 Pattern of relapse will be evaluated by number of patients with patterns of tumor recurrence such as local recurrence, marginal recurrence, regional recurrence, distant metastasis, and second primary tumor divided by the total number of evaluable patients. Exact binomial 95% confidence interval for the point estimate will be provided.
  - 16.3.2.5.1 Local tumor recurrence is defined as any tumor recurrence inside the CTV.
  - 16.3.2.5.2 Marginal tumor recurrence is defined as any tumor recurrence beyond the CTV to within a 3 cm distance from the edge of the CTV.
  - 16.3.2.5.3 Distant tumor recurrence is defined as any tumor that develops distantly from the primary site of sarcoma.

- 16.3.2.5.4 Second primary tumor is defined as any different histology of sarcoma or any other type of malignancy inside or outside the radiation field.
- 16.3.2.6 Adverse Events: All eligible patients that have initiated treatment will be considered evaluable for assessing adverse event rate(s). The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Late toxicities (as defined in sections 16.3.2.4) will be summarized separately.
- 16.3.2.7 Quality of Life Measurements PROMIS-10: Results from the ten-item PROMIS questionnaire will be used to evaluate physical health and mental health, separately. Changes in raw score from baseline to 24-months post-surgery will be assessed, in each of the physical and mental health domains. The Wilcoxon signed-rank test will be utilized to assess changes in raw PROMIS scores. Mean change, along with standard deviation will be reported.

A scoring table to compare this patient population to global means may be utilized for various timepoints. However, because this scoring table is prepared for a fixed set of items, it can only be used when an examinee responds to all of the items in the set. This, along with all other analyses, including graphical representations and comparisons between other timepoints or subgroups of patients may be performed, but will be considered exploratory.

16.3.2.8 Quality of Life Measurements – TESS: Results from the Toronto Extremity Salvage Score (TESS) questionnaire will be used to evaluate functional outcomes. The TESS specifically measures performance of activities of daily living, and is separated into upper and lower extremity versions (29 and 30 questions, respectively).

Patients will fill out the appropriate version, and point totals will be summed. Mean change from baseline to 24 months post-surgery, along with standard deviation will be reported by version. The Wilcoxon signed-rank test will be used to assess changes in TESS scores within questionnaires. All other analyses, including graphical representations, GEE model creation, and comparisons between different timepoints or subgroups of patients may be performed, but will be considered exploratory.

#### 16.4 Data Safety and Monitoring

- 16.4.1 Safety Review: The principal investigator(s) and the study statistician will review the study monthly to identify accrual, adverse event, and any endpoint problems that might be developing. The Mayo Clinic Cancer Center (MCCC) Data Safety Monitoring Board (DSMB) is responsible for reviewing accrual and safety data for this trial at least biannually, based on reports provided by the MCCC Statistical Office.
- 16.4.2 Adverse Event Stopping Rules: The stopping rule specified below is based on the knowledge available at study development. We note that the Adverse Event Stopping Rule may be adjusted in the event of either (1) the study re-opening to accrual or (2) at any time during the conduct of the trial and in consideration of newly acquired information regarding the adverse event profile of the treatment(s) under investigation. The study team may choose to suspend accrual because of unexpected adverse event profiles that have not crossed the specified rule below.

Accrual may be temporarily suspended to this study if at any time we observe events considered at least possibly related to Radiation Therapy (i.e., an adverse event with attribute specified as "possible", "probable", or "definite") that satisfy one of the following:

- If 8 or more of the first 20 patients (or 40% or more of all patients after 10 are accrued) experience a Grade 3+ AE.
- If 4 or more experience a Grade 5 AE at any time.

After consideration by the study team (Study Chair, statistician, etc.), a decision will be made as to whether accrual can be resumed. In addition, we will review grade 4 and 5 adverse events deemed "unrelated" or "unlikely to be related", to verify their attribution and to monitor the emergence of a previously unrecognized treatment-related adverse event.

#### 16.5 Subset Analyses for Minorities

#### 16.5.1 Study Availability

This study will be available to all eligible patients, regardless of gender, race or ethnic origin.

#### 16.5.2 Statistical Analysis by Subset

There is no information currently available regarding differential effects of this radiation treatment in subsets defined by race, gender, or ethnicity, and there is no reason to expect such differences to exist. Therefore, although the planned analyses will look for differences in treatment effect based on racial groupings, the sample size is not increased in order to provide additional power for subset analyses.

MC1973

#### 16.5.3 Regional Population

The geographical region served by MCCC has a population which includes approximately 10% minorities. Expected sizes of racial by gender subsets are shown in the following table:

| Accrual Targets | | | |
|-------------------------------------------|------------|-------|-------|
| | Sex/Gender | | |
| Ethnic Category | Females | Males | Total |
| Hispanic or Latino | 3 | 3 | 6 |
| Not Hispanic or Latino | 57 | 57 | 114 |
| Ethnic Category: Total of all subjects* | 60 | 60 | 120 |
| Racial Category | | | |
| American Indian or Alaskan Native | 2 | 1 | 3 |
| Asian | 1 | 2 | 3 |
| Black or African American | 2 | 2 | 4 |
| Native Hawaiian or other Pacific Islander | 1 | 1 | 2 |
| White | 54 | 54 | 108 |
| Racial Category: Total of all subjects* | 60 | 60 | 120 |

Ethnic Categories:

**Hispanic or Latino** – a person of Cuban, Mexican, Puerto Rican, South or Central American, or other Spanish culture or origin, regardless of race. The term "Spanish origin" can also be used in addition to "Hispanic or Latino."

#### **Not Hispanic or Latino**

Racial Categories:

American Indian or Alaskan Native – a person having origins in any of the original peoples of North, Central, or South America, and who maintains tribal affiliations or community attachment.

Asian – a person having origins in any of the original peoples of the Far East, Southeast Asia, or the Indian subcontinent including, for example, Cambodia, China, India, Japan, Korea, Malaysia, Pakistan, the Philippine Islands, Thailand, and Vietnam. (Note: Individuals from the Philippine Islands have been recorded as Pacific Islanders in previous data collection strategies.)

Black or African American – a person having origins in any of the black racial groups of Africa. Terms such as "Haitian" or "Negro" can be used in addition to "Black or African American."

Native Hawaiian or other Pacific Islander – a person having origins in any of the original peoples of Hawaii, Guam, Samoa, or other Pacific Islands.

White – a person having origins in any of the original peoples of Europe, the Middle East, or North Africa.

#### 17.0 Pathology Considerations/Tissue Biospecimens

N/A

#### 18.0 Records and Data Collection Procedures

#### 18.1 Data Collection and Processing

All data will be entered into electronic case report forms (eCRF's) through the Medidata Rave system. Case report forms will be automatically rolled out based on a predetermined, and visit based schedule to improve study staff workflow and data quality. Data will be exported nightly to a secure FTP for analysis and reporting.

#### 18.2 Data Security and Confidentiality

The Medidata Rave database access model is role based and fully auditable at the study, form, and field levels. Data will be de-identified whenever possible and the ability to update will be limited to necessary staff. Access will be managed by the Mayo CTMS Service and Solution Center, under a controlled and monitored access request system. Medidata's platform specifically supports Electronic Record and Electronic Signature (ER/ES) requirements, including US 21 CFR part 11.

#### 18.3 Data Quality Assurance

Each eCRF will contain edit checks and custom functions to ensure the highest possible data quality. Only necessary eCRF's will be available for data entry to reduce the possibility of erroneous entry.

The edit checks and custom functions on the eCRF's will trigger queries requesting the attention of appropriate study staff. The fields will be marked in pink to allow study staff to quickly identify the data fields that require attention or actions. Additionally, secure email notifications will be sent for adverse event tracking and monitoring.

#### 19.0 Budget

- 19.1 Costs charged to patient: Routine clinical care
- 19.2 Tests to be research funded: None

#### 20.0 References

- 1. Rosenberg SA, Tepper J, Glatstein E, et al. The treatment of soft-tissue sarcomas of the extremities: prospective randomized evaluations of (1) limb-sparing surgery plus radiation therapy compared with amputation and (2) the role of adjuvant chemotherapy. Ann Surg 1982;196:305-15.
- 2. Pisters PW, Harrison LB, Leung DH, Woodruff JM, Casper ES, Brennan MF. Long-term results of a prospective randomized trial of adjuvant brachytherapy in soft tissue sarcoma. J Clin Oncol 1996;14:859-68.
- 3. Yang JC, Chang AE, Baker AR, et al. Randomized prospective study of the benefit of adjuvant radiation therapy in the treatment of soft tissue sarcomas of the extremity. J Clin Oncol 1998:16:197-203.
- 4. Barkley HT, Jr., Martin RG, Romsdahl MM, Lindberg R, Zagars GK. Treatment of soft tissue sarcomas by preoperative irradiation and conservative surgical resection. Int J Radiat Oncol Biol Phys 1988;14:693-9.
- 5. Lindberg RD, Martin RG, Romsdahl MM, Barkley HT, Jr. Conservative surgery and postoperative radiotherapy in 300 adults with soft-tissue sarcomas. Cancer 1981;47:2391-7.
- 6. O'Sullivan B, Davis AM, Turcotte R, et al. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet 2002;359:2235-41.
- 7. Beane JD, Yang JC, White D, Steinberg SM, Rosenberg SA, Rudloff U. Efficacy of adjuvant radiation therapy in the treatment of soft tissue sarcoma of the extremity: 20-year follow-up of a randomized prospective trial. Ann Surg Oncol 2014;21:2484-9.
- 8. Cannon CP, Ballo MT, Zagars GK, et al. Complications of combined modality treatment of primary lower extremity soft-tissue sarcomas. Cancer 2006;107:2455-61.
- 9. DeLaney TF, Spiro IJ, Suit HD, et al. Neoadjuvant chemotherapy and radiotherapy for large extremity soft-tissue sarcomas. Int J Radiat Oncol Biol Phys 2003;56:1117-27.
- 10. Moore J, Isler M, Barry J, Mottard S. Major wound complication risk factors following soft tissue sarcoma resection. Eur J Surg Oncol 2014;40:1671-6.
- 11. Wang D, Zhang Q, Eisenberg BL, et al. Significant Reduction of Late Toxicities in Patients With Extremity Sarcoma Treated With Image-Guided Radiation Therapy to a Reduced Target Volume: Results of Radiation Therapy Oncology Group RTOG-0630 Trial. J Clin Oncol 2015;33:2231-8.
- 12. Scharschmidt T, Chen Y, Wand D, Chi Y, Kayton M, J S. ARST1321: Pazopanib neoadjuvant trial in non-rhabdomysarcoma soft tissue sarcomas: A report of major wound complications. J Clin Oncol 2019;37.
- 13. Davis AM, O'Sullivan B, Bell RS, et al. Function and health status outcomes in a randomized trial comparing preoperative and postoperative radiotherapy in extremity soft tissue sarcoma. J Clin Oncol 2002;20:4472-7.
- 14. Davis AM, O'Sullivan B, Turcotte R, et al. Late radiation morbidity following randomization to preoperative versus postoperative radiotherapy in extremity soft tissue sarcoma. Radiother Oncol 2005;75:48-53.
- 15. Davis AM, Sennik S, Griffin AM, et al. Predictors of functional outcomes following limb salvage surgery for lower-extremity soft tissue sarcoma. J Surg Oncol 2000;73:206-11.
- 16. Haas RL, Delaney TF, O'Sullivan B, et al. Radiotherapy for management of extremity soft tissue sarcomas: why, when, and where? Int J Radiat Oncol Biol Phys 2012;84:572-80.

- 17. Haas RL, Miah AB, LePechoux C, et al. Preoperative radiotherapy for extremity soft tissue sarcoma; past, present and future perspectives on dose fractionation regimens and combined modality strategies. Radiother Oncol 2016;119:14-21.
- 18. Dearnaley D, Syndikus I, Mossop H, et al. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol 2016;17:1047-60.
- 19. Haviland JS, Owen JR, Dewar JA, et al. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol 2013;14:1086-94.
- 20. Whelan TJ, Pignol JP, Levine MN, et al. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med 2010;362:513-20.
- 21. Kosela-Paterczyk H, Szacht M, Morysinski T, et al. Preoperative hypofractionated radiotherapy in the treatment of localized soft tissue sarcomas. Eur J Surg Oncol 2014;40:1641-7.
- 22. Pennington JD, Eilber FC, Eilber FR, et al. Long-term Outcomes With Ifosfamide-based Hypofractionated Preoperative Chemoradiotherapy for Extremity Soft Tissue Sarcomas. Am J Clin Oncol 2018;41:1154-61.

## **Appendix I ECOG Performance Status**

| ECOG PERFORMANCE STATUS* | |
|---|---|
| Grade | ECOG |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair. |
| 5 | Dead |

<sup>\*</sup>As published in Am. J. Clin. Oncol.:

Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982.

The ECOG Performance Status is in the public domain therefore available for public use. To duplicate the scale, please cite the reference above and credit the Eastern Cooperative Oncology Group, Robert Comis M.D., Group Chair.

From http://www.ecog.org/general/perf stat.html

# Appendix II – PROMIS-10

# **Mayo Patient Survey**

Survey Date: \_\_\_\_\_ mm/dd/yyyy

| Please respond to each item by choosing one numb | er per | ro | w. | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Excelle | Very | | Good | Fair | Poor |
| In general, would you say your <b>health</b> is: | | | 0 | 0 | | 0 | 0 | 0 |
| in general, would you say your nearth is. | | | 5 | 4 | | 3 | 2 | 1 |
| In general, would you say your quality of life is: | | | 0 | 0 | | 0 | 0 | 0 |
| in general, media yea say year <b>quarry or me</b> is. | | | 5 | 4 | | 3 | 2 | 1 |
| In general, how would you rate your physical health? | | | 0 | 0 | | 0 | C | 0 |
| | | | 5 | 4 | | 3 | 2 | 1 |
| In general, how would you rate your mental health, including | | | 0 | 0 | | 0 | 0 | 0 |
| your mood and your ability to think? | | | 5 | 4 | | 3 | 2 | 1 |
| In general, how would you rate your satisfaction with your | | | 0 | 0 | | 0 | 0 | 0 |
| social activities and relationships? | | | 5 | 4 | | 3 | 2 | 1 |
| In general, please rate how well you carry out your usual | | | 0 | 0 | | 0 | 0 | 0 |
| social activities and roles. (Includes activities at home, work, community, parenting, marriage, friends.) | | | 5 | 4 | | 3 | 2 | 1 |
| | | Co | mpletely | Mostly | / М | oderately | A<br>little | Not at all |
| To what extent are you able to carry out your everyday physical | | | 0 | 0 | | 0 | 0 | 0 |
| activities such as walking,climbing stairs carrying groceries, or moving a chair? | | | 5 | 4 | | 3 | 2 | 1 |
| In the past 7 days | | | | | | | | |
| | | | Never | Rarely | Sor | netimes | Often | Always |
| How often have you been bothered by emotional problems such | | | 0 | 0 | | 0 | 0 | 0 |
| as feeling anxious, depressed or irritable? | | | 1 | 2 | | 3 | 4 | 5 |
| | | | None | Mild | Mo | derate | Severe | Very Severe |
| How would you rate your fatique on average? | | | 0 | 0 | | 0 | 0 | 0 |
| now would you rate your ranger on average: | | | 1 | 2 | | 3 | 4 | 5 |
| | No<br>pain | 0 | _ | 0 0 | , | 0.0 | 0 ( | Wors<br>imaginab |
| How would you rate your <b>pain</b> on average? | 0 | 1 | 2 | 3 4 | | 5 6 | 7 8 | |

# **Appendix III- TESS**

| Radiation Therapy Oncology Group Phase II Soft Tissue Sarcoma Toronto Extremity Salvage Score (TESS) | RTOG Study 0830 Case # PLACE LABEL HERE |
|---|---|
| | Institution No. |
| | Participant's Initials Participant's I.D. No. |
| AMENDED DATA YES INSTRUCTIONS: This sheet is questionnaire. This page must be physician, etc.) See detailed instru | s the cover page used for submission of the (TESS) completed by the medical staff (nurse, data manager, uctions for TESS questionnaire. |
| 1 LITIME POINT(1) 1 Baseline 2 12 months from start of treatment | 4 SPECIFY METHOD OF COMPLETION(7) 0 Not applicable (not completed) 1 At appointment |
| 3 18 months from start of treatment<br>4 24 months from start of treatment | 2 By mail<br>3 By telephone<br>9 Unknown |
| 2 WAS PATIENT QUESTIONNAIRE COMPLETED?(2) 1 No (Skip to question 3) | 6 DID THE PATIENT REQUIRE ANY ASSISTANCE IN COMPLETING THE QUESTIONNAIRE?(II) |
| 2 Yes 2A DATE PATIENT QUESTIONNAIRE COMPLETED | Not applicable (not completed) No Yes Unknown if assistance was given |
| | 8 SPECIFY THE PERSON WHO ASSISTED THE PATIENT(R) |
| REASON QUESTIONNAIRE WAS NOT COMPLETED(4) O Not applicable, questionnaire was completed 1 Patient refused due to lilness 2 Patient refused for other reason, specify | 0 Not applicable (not completed, no assistance) 1 Staff member 2 Family 3 Other, specify |
| Signature of person completing this form(%) | Date form completed(15) |
| The state of the s | January Compression (iii) |



Radiation Therapy Oncology Group Phase II Soft Tissue Sarcoma Toronto Extremity Salvage Score (TESS) RTOG 8tudy 0830

Case #

PLACE LABEL HERE

Institution Participant's Initials Institution No. Participant's I.D. No.

# Toronto Extremity Salvage Score (TESS) Administration of the Questionnaire

51

#### General Guidelines

This questionnaire is designed as a measure of physical disability for patients undergoing limb salvage surgery for musculoskeletal tumours. It is a self-administered questionnaire.

There is an upper extremity and lower extremity version of the questionnaire. It is recommended that study personal complete the general information and review the instructions and sample questions with the subjects. The subjects can independently answer the remaining questions. Total completion time of the questionnaire averages 10 minutes.

#### Scoring

Each question is a measure of the difficulty that the individual has performing the task. The total potential score for an item is a perfect performance score (ie. 5).

The scale has been designed to allow individuals to respond to a nonapplicable category on an item if it is not something they perform in their everyday life. Consequently, a total questionnaire score, if desired, would be a standardized score ranging from 0 to 100 calculated by:

> sum of the item scores - # items X 100%, possible score range

where, sum of the item scores = sum of difficulty responses # items = items completed excluding the NA repsonse items possible score range = (5 x #items) - (1 x #items)

#### Mail Administration

The TESS questionnaires have been administered by mail and, although formal testing of measurement properties has not been undertaken, patients are able and willing to complete the forms and the scores fall within anticipated ranges.

| SS | RTOG 8tudy 0830 | Case # |
|---|---|---|
| | PLACE I | ABEL HERE |
| | Institution | Institution No. |
| | Participant's Initials | Partiolpant's I.D. No. |
| Toronto Extremity Salvage Score (Davis, 1996) Upper Extremity Questionnaire | | |
| Completed by patient at baseline, 12, 18, 18, 19 | | |
| TESS - UPF | PER EXTREMITY | |
| Patient Study ID#: Patie | nt initials:<br>(first/middle/last) | |
| | Completion Date: (day/monti | n/year) |
| Months from start of treatment Baseline 12 months 18 months 24 months | | |
| Site: 1 Bone Side | of Lesion: 1Right | |
| 2 Soft Tissue | 2Left | |
| Are you: 1right handed 2left handed | | |
| The following questions are about activities commonly p<br>asks that you mark each item (as in the examples below<br>to perform each task during the <u>past week.</u> Some act<br>extremely difficult or impossible. | w) opposite the description the | at best describes your ability |

| _ | | | |
|---|---|---|---|
| SS | | RTOG Study 0830 | Case # |
| | | PLACE LABEL HERE | |
| | | Institution | Institution No. |
| | | Participant's Initials | Partiolpant's I.D. No. |
| | EVANDI E | | |
| | EXAMPLE Decline venetables in: | | |
| | Peeling vegetables is: 1impossible to do. | | |
| | 2extremely difficult. | | |
| | 3moderately difficult. | | |
| | 4 a little bit difficult. | • | |
| | 5 not at all difficult. | | |
| | onat all allique. | | |
| | 888This task is not ap | plicable for me. | |
| | You should choose the response "Impossible to do" if | the activity is something that yo | u normally do in your |
| | daily activities but are now unable to do because of physi | ical limitations such as weakness | stiffness or pain. |
| | If you do not perform an activity as part of your normal life | estyle you would choose the resp | onse "888" to Indicate |
| | that the Item is not applicable. | | |
| | Mark all Items ensuring that you choose the description t | hat most accurately describes yo | ur abilities in the <u>past</u> |
| | week. | | |
| | The following questions ask about your ability to perform | activities that are common to eve | ryday life. Considering |
| | the amount of difficulty you have performing the activity d | ue to the current problem you are | having with your arm, |
| | please answer the questions by choosing the answer that | it best describes your ability to d | o the activity over the |
| | past week. | | |
| | 1) Putting on a pair of pants is: | | |
| | 1impossible to do. | | |
| | 2extremely difficult. | | |
| | <ol> <li>moderately difficult.</li> </ol> | | |
| | 4a little bit difficult. | | |
| | 5not at all difficult. | ellechie des es | |
| | 888This task is not ap | plicable for me. | |
| | 2) Tying shoe laces is: | | |
| | 1impossible to do. | | |
| | 2extremely difficult. | | |
| | <ol> <li>moderately difficult.</li> <li>a little bit difficult.</li> </ol> | | |
| | 4a little bit difficult. 5not at all difficult. | | |
| | 5not at an difficult. | | |
| | 888This task is not ap | nlicable for me | |
| | This task is not ap | providente nut tiffe. | |

| SS | | RTOG Study 0830 | Case # |
|---|---|---|---|
| | | PLACE LAB | EL HERE |
| | | Institution | Institution No. |
| | | Participant's Initials | Participant's I.D. No. |
| | 3) Putting on socks or stockings is: | | |
| | 4 | _ | |
| | 1impossible to d<br>2extremely diffic | | |
| | 3moderately diff | | |
| | 4a little bit difficu | | |
| | 5not at all difficu | lt. | |
| | 888This task is no | t applicable for me. | |
| | 4) Showering is: | | |
| | 1impossible to d | o. | |
| | 2extremely diffic | ult. | |
| | 3moderately diffi | icult. | |
| | 4a little bit difficu | | |
| | 5not at all difficu | lt. | |
| | 888This task is no | t applicable for me. | |
| | 5) Dressing my arms and upper body is: | | |
| | 1impossible to d | o. | |
| | 2extremely diffic | | |
| | 3moderately diff | | |
| | 4a little bit difficu | | |
| | 5not at all difficu | it. | |
| | 888This task is no | t applicable for me. | |
| | 6) Buttoning a shirt is: | | |
| | 1impossible to d | o. | |
| | 2extremely diffic | ult. | |
| | 3moderately diff | | |
| | 4a little bit difficu | | |
| | 5not at all difficu | lt. | |
| | 888 This task is no | t applicable for me. | |
| | | 0630 | SS 03-25-08 5 of 21 |

| 66 | RTOG Study 0830 | Case # |
|---|---|---|
| 55 | DIACETA | BEL HERE |
| | FLACE LA | ADEL HERE |
| | Institution | Institution No. |
| | Participant's Initials | Partiolpant's I.D. No. |
| 7) Tying a tie or a bow at the neck of a blouse is: | | |
| 1Impossible to | | |
| 2exfremely diffi | | |
| 3moderately df | | |
| 4a little bit diffic | | |
| 5not at all diffic | sult. | |
| 888This task is n | ot applicable for me. | |
| 8) Buillian an araba un anabardan la | | |
| 8) Putting on make-up or shaving is: | | |
| 1Impossible to | | |
| 2extremely diffi | | |
| 3moderately di | | |
| 4a little bit diffic<br>5not at all diffic | | |
| bnot at all dillo | uii. | |
| 888This task is n | ot applicable for me. | |
| 9) Brushing your teeth is: | | |
| 1Impossible to | do. | |
| 2extremely diffi | lcult. | |
| 3moderately df | fficult. | |
| 4a little bit diffic | cult. | |
| 6not at all diffic | eult. | |
| 888 This task is n | ot applicable for me. | |
| 0001185 task ts 11 | ot applicable for file. | |
| 10) Brushing your hair is: | | |
| 1impossible to | do. | |
| 2exiremely diffi | | |
| 3moderately di | | |
| 4a little bit diffic | | |
| 5not at all diffic | | |
| 888This task is n | | |

0630 SS 03-25-08 6 of 21

| SS | RTOG Study 0830 | Case # |
|---|---|---|
| | PLACE LAB | EL HERE |
| | Institution | teeds dree to |
| | Participant's initials | Institution No. Partiolpant's I.D. No. |
| 11) Doing light household chores is: | | |
| 1impossible to do | | |
| 2extremely difficu<br>3moderately diffic | | |
| 3moderately diffic<br>4a little bit difficult | | |
| 5not at all difficult | | |
| 0not at all direction | • | |
| 888This task is not | applicable for me. | |
| 12) Gardening or yard work is: | | |
| 1impossible to do | ı. | |
| 2extremely difficu | | |
| 3moderately diffic | | |
| 4a little bit difficult | L. | |
| 5not at all difficult | L | |
| 888This task is not | applicable for me. | |
| 13) Preparing and serving meals is: | | |
| 1impossible to do | | |
| 2extremely difficu | | |
| 3moderately diffic | | |
| 4a little bit difficult | | |
| 5not at all difficult | | |
| 888This task is not | applicable for me. | |
| 14) Cutting food while eating is: | | |
| 1impossible to do | L. | |
| 2extremely difficu | lt. | |
| 3moderately diffic | zult. | |
| 4a little bit difficult | t. | |
| 5not at all difficult | L | |
| 888This task is not | applicable for me. | |

| | | | (nrong plantagener | |
|---|---|---|---|---|
| SS | | | RTOG Study 0830 | Case # |
| | | | PLACE LAB | EL HERE |
| | | | Institution | Institution No. |
| | | | Participant's Initials | Participant's I.D. No. |
| | 15) Drinking from a glass is: | | | |
| | 10) Dilliking from a glass is. | 1impossible to d | to. | |
| | | 2extremely diffic | | |
| | | 3moderately diff | | |
| | | 4 a little bit diffici | | |
| | | 5not at all difficu | ult. | |
| | 8 | 388This task is no | ot applicable for me. | |
| | 16) Performing heavy househ | iold chores is: | | |
| | | 1impossible to d | do. | |
| | | 2extremely diffic | | |
| | | 3moderately diff | | |
| | | 4a little bit diffic | | |
| | | 5not at all difficu | ult. | |
| | 8 | 388This task is no | ot applicable for me. | |
| | 17) Going shopping is: | | | |
| | | 1impossible to d | <b>1</b> 0. | |
| | | 2extremely diffic | cult. | |
| | | 3moderately diff | fleuit. | |
| | | 4a little bit diffici | ult. | |
| | | 5not at all difficu | ult. | |
| | 8 | 388This task is no | ot applicable for me. | |
| | 18) Giving or receiving chang | je (le. colns or bills) l | 5: | |
| | | 1impossible to d | <b>1</b> 0. | |
| | | 2extremely diffic | cult. | |
| | | 3moderately diff | flouit. | |
| | | 4a little bit diffici | ult. | |
| | | 5not at all difficu | ult. | |
| | 8 | 888This task is no | ot applicable for me. | |

| SS | | RTOG Study 0630 | Case # |
|---|---|---|---|
| | | PLACE LAB | EL HERE |
| | | Institution | Institution No. |
| | | Participant's Initials | Participant's I.D. No. |
| | 19) Carrying a shopping bag or briefcase is: | | |
| | 1impossible to | do. | |
| | 2extremely diff | | |
| | _ | | |
| | 4a little bit diffic | | |
| | 6not at all diffic | zult. | |
| | 888This task is n | ot applicable for me. | |
| | 20) Lifting a box to an overhead shelf is: 1impossible to | do | |
| | 2extremely diff | | |
| | 3moderately di | | |
| | 4 a little bit diffic | | |
| | 5not at all diffic | cult. | |
| | 888This task is n | ot applicable for me. | |
| | 21) Turning a key in a lock is: | | |
| | 1impossible to | | |
| | 2extremely diff | | |
| | 3moderately di<br>4a little bit diffic | | |
| | 4a little bit diffic<br>5not at all diffic | | |
| | 5ilot at all dillo | un. | |
| | 888This task is n | not applicable for me. | |
| | 22) Pushing or pulling open a door is: | | |
| | 1impossible to | | |
| | 2extremely diff | | |
| | 3moderately di<br>4a little bit diffic | | |
| | 4a nut at all diffic | | |
| | 5noratan dine | MI. | |
| | 888This task is n | not applicable for me. | |

| SS | | RTOG Study 0830 | Case # |
|---|---|---|---|
| | | PLACE LAB | EL HERE |
| | | Institution | Institution No. |
| | | Participant's Initials | Participant's I.D. No. |
| | 23) Writing is: | | |
| | 1impossible to do. 2extremely difficult. | | |
| | 3moderately difficul | | |
| | 4a little bit difficult. | - | |
| | 5 not at all difficult. | | |
| | 888This task is not a | pplicable for me. | |
| | 24) Picking up small items is: | | |
| | 1impossible to do. | | |
| | 2extremely difficult. | | |
| | 3moderately difficul | t. | |
| | 4a little bit difficult. 5not at all difficult. | | |
| | bnot at all difficult. | | |
| | 888This task is not a | pplicable for me. | |
| | 25) Completing my usual duties at work is: (Work incl | udes a job outside the home or as | a homemaker.) |
| | 1impossible to do. | • | • |
| | 2extremely difficult. | | |
| | 3moderately difficul | it. | |
| | 4a little bit difficult. | | |
| | 5not at all difficult. | | |
| | 888This task is not a | pplicable for me. | |
| | 26) Working my usual number of hours is: (Work homemaker.) | king includes both a job outside | the home and as a |
| | 1impossible to do. | | |
| | 2extremely difficult. | | |
| | 3moderately difficul | | |
| | 4a little bit difficult. | | |
| | 5not at all difficult. | | |
| | 888This task is not a | pplicable for me. | |
| | | | , |

| SS | | RTOG Study 0830 | Case # |
|---|---|---|---|
| | | PLACE LAB | EL HERE |
| | | Institution | Institution No. |
| | | Participant's initials | Participant's I.D. No. |
| | 27) Participating in my usual leisure activities is: | | |
| | 1impossible to do | | |
| | 2extremely difficu | | |
| | 3moderately diffic | | |
| | 4a little bit difficult | | |
| | 5not at all difficult | | |
| | 888This task is not | applicable for me. | |
| | 28) Socializing with friends and family is: | | |
| | 1impossible to do | | |
| | 2extremely difficu | | |
| | 3moderately diffic | | |
| | 4a little bit difficult | | |
| | 5not at all difficult | | |
| | 888This task is not | applicable for me. | |
| | 29) Participating in my usual sporting activities is: | | |
| | 1impossible to do | | |
| | 2extremely difficu | It. | |
| | 3moderately diffic | ult. | |
| | 4a little bit difficult | | |
| | 5not at all difficult | | |
| | 888This task is not | applicable for me. | |
| | 1) Considering all the activities in which I participa | ate in daily life, I would rate my | ability to perform these |
| | activities during the past week as: | | |
| | 1Impossible to d | | |
| | 2extremely diffic | | |
| | 3moderately diff | | |
| | 4a little bit diffici | | |
| | 5not at all difficu | ult. | |

| 18.31 I | | RTOG Study 0630 | Case # |
|---|---|---|---|
| | | PLACE I | ABEL HERE |
| | | Institution | Institution No. |
| | | Participant's initials | Partiolpant's I.D. No. |
| 2) I would rate myself a | se halna : | | |
| 2) I would rate myself a | is being . | | |
| | 1completely disal | bled | |
| | 2severely disable | d. | |
| | 3moderately disa | bled. | |
| | 4mildly disabled. | | |
| | 5not at all disable | d. | |
| | on any activities you find difficu | | |
| | urrently have in your arm that y | you feel are important and ha | eve not been asked about in |
| this questionnaire. | | | |
| Please check to make s | sure that you have not missed | I any questions. | |
| Please check to make s | sure that you have not missed | I any questions. | |
| | sure that you have not missed<br>e time to answer these questi | | |

# Radiation Therapy Oncology Group Phase II Soft Tissue Sarcoma Toronto Extremity Salvage Score (TESS)

RTOG Study 0830

Case #

#### PLACE LABEL HERE

Institution Participant's initials Institution No.
Participant's I.D. No

| | TESS - LOWER EXTREMITY | |
|---|---|---|
| Patient Study ID#: | Patient Initials: | |
| | (first/middle/last) | |
| Date of birth: | Form Completion Date: | |
| (day/month/year) | (day/month/year) | |
| Months from start of treatment | Baseline | |
| World is from start or freatment | 12 months | |
| | 18 months | |
| | 24 months | |
| Site: 1 Bone | | |
| 2 Soft Tissue | | |
| The following questions are about ac | ivities commonly performed in daily life. Each question | |
| 9 1 | | |
| asks that you mark each item (as in | he examples below) apposite the description that heat d | learnings your shility |
| | he examples below) opposite the description that best of | |
| to perform each task during the pas | he examples below) opposite the description that best of<br>twook. Some activities will be extremely easy for you | |
| to perform each task during the pas | | |
| to perform each task during the pas<br>extremely difficult or impossible. | | |
| to perform each task during the pas<br>extremely difficult or impossible. | | |
| to perform each task during the <u>pas</u><br>extremely difficult or impossible.<br><b>EXAMPLE</b><br>Riding a bicycle is: | wook. Some activities will be extremely easy for you | |
| to perform each task during the <u>pas</u><br>extremely difficult or impossible.<br>EXAMPLE<br>Riding a bicycle is: | twook. Some activities will be extremely easy for you impossible to do. | |
| to perform each task during the <u>pas</u><br>extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | wook. Some activities will be extremely easy for you<br>impossible to do.<br>extremely difficult. | |
| to perform each task during the pase<br>extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | impossible to doextremely difficult. | |
| to perform each task during the <u>pas</u><br>extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | impossible to doextremely difficulta little bit difficult. | |
| to perform each task during the pase<br>extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | impossible to doextremely difficult. | |
| to perform each task during the <u>pass</u> extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 2 3 4 | impossible to doextremely difficulta little bit difficult. | |
| to perform each task during the pase extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | _impossible to doextremely difficultnoderately difficultnot at all difficultThis task is not applicable for me. | to do, others will be |
| to perform each task during the pase extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | impossible to doextremely difficultmoderately difficultnot at all difficultThis task is not applicable for me. possible to do" if the activity is something that you in | normally do in your |
| to perform each task during the pase extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | _impossible to doextremely difficultnoderately difficultnot at all difficultThis task is not applicable for me. | normally do in your |
| to perform each task during the pase extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | impossible to do. extremely difficult. moderately difficult. a little bit difficult. not at all difficult. This task is not applicable for me. possible to do" if the activity is something that your do because of physical limitations such as weakness, si | normally do in your tiffness or pain. |
| to perform each task during the pass extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | impossible to doextremely difficultmoderately difficultnot at all difficultThis task is not applicable for me. possible to do" if the activity is something that you in | normally do in your tiffness or pain. |
| to perform each task during the pass extremely difficult or impossible. EXAMPLE Riding a bicycle is: 1 | impossible to do. extremely difficult. moderately difficult. a little bit difficult. not at all difficult. This task is not applicable for me. possible to do" if the activity is something that your do because of physical limitations such as weakness, si | normally do in your<br>tiffness or pain. |

| SS | RTOG 8 tudy 0830 | Case # |
|---|---|---|
| | PLACE | LABEL HERE |
| | Institution | Institution No. |
| | Participant's initials | Institution No. Participant's I.D. No. |
| The following questions ask about your ability to perform | | |
| the amount of difficulty you have performing the activity | | |
| please answer the questions by choosing the answer t | that best describes your ability | to do the activity over the |
| past week. | | |
| 1) Putting on a pair of pants is: | | |
| 1impossible to do. | | |
| 2extremely difficul | | |
| 3moderately diffice<br>4a little bit difficult | | |
| 5not at all difficult. | | |
| onos se un comode. | | |
| 888This task is not a | applicable for me. | |
| 2) Putting on shoes is: | | |
| 1impossible to do. | | |
| 2extremely difficul | t. | |
| 3moderately diffic | | |
| 4a little bit difficult | | |
| 5not at all difficult. | | |
| 888This task is not a | applicable for me. | |
| 3) Putting on socks or stockings is: | | |
| 1impossible to do. | | |
| 2extremely difficul | | |
| 3moderately diffic | ult. | |
| 4a little bit difficult | | |
| 5not at all difficult. | | |
| 888This task is not a | applicable for me. | |
| 4) Showering is: | | |
| 1impossible to do. | | |
| 2extremely difficul | | |
| 3moderately diffic | ult. | |
| 4a little bit difficult | | |
| 5not at all difficult. | | |
| 888This task is not a | applicable for me. | |

| SS | RTOG Study 083 | 0 Case # |
|---|---|---|
| 00 | PL | ACE LABEL HERE |
| | Institution | Institution No. |
| | Participant's init | |
| 5) Light household chores suc | th as tidying and dusting are:<br>1impossible to do. | |
| | 2extremely difficult. | |
| | 3moderately difficult. | |
| | 4a little bit difficult. | |
| | 5not at all difficult. | |
| 8 | 38This task is not applicable for me. | |
| 6) Gardening and yard work a | · •: | |
| | 1impossible to do. | |
| | 2extremely difficult. | |
| | 3moderately difficult. | |
| | 4a little bit difficult. | |
| | 5not at all difficult. | |
| 8 | 88This task is not applicable for me. | |
| 7) Preparing and serving meal | s is: | |
| | 1impossible to do. | |
| | 2extremely difficult. | |
| | <ol> <li>moderately difficult.</li> </ol> | |
| | 4a little bit difficult. | |
| | 5not at all difficult. | |
| 8 | 38This task is not applicable for me. | |
| 8) Going shopping is: | | |
| | 1impossible to do. | |
| | 2extremely difficult. | |
| | 3moderately difficult. | |
| | 4a little bit difficult. | |
| | 5not at all difficult. | |
| 8 | 38This task is not applicable for me. | |
| ( | | |

| SS | | RTOG Study 0830 | Case # |
|---|---|---|---|
| | | PLACE | LABEL HERE |
| | | Institution | Institution No. |
| | | Participant's Initials | Partiolpant's I.D. No. |
| 9) Heavy household chore | s such as vacuumin | n and moving furniture is: | |
| o) neavy nousehold choic | 1impossible | _ | |
| | 2extremely of | | |
| | 3moderately | | |
| | 4a little bit di | fficult. | |
| | 5not at all di | fficult. | |
| | 888This task it | s not applicable for me. | |
| 10) Getting in and out of the | ne bath tub Is: | | |
| | 1Impossible | | |
| | 2extremely o | | |
| | 3moderately | | |
| | 4a little bit di | | |
| | 5not at all di | mcurt. | |
| | 888This task is | s not applicable for me. | |
| 11) Getting out of bed is: | | | |
| | 1Impossible | to do. | |
| | 2extremely of | imcuit. | |
| | 3moderately | difficult. | |
| | 4a little bit di | | |
| | 5not at all dit | Mcult. | |
| | 888This task is | s not applicable for me. | |
| 12) Rising from a chair is: | | | |
| , | 1impossible | to do. | |
| | 2extremely of | imcult. | |
| | 3moderately | difficult. | |
| | 4a little bit di | ifficult. | |
| | 5not at all di | Moult. | |
| | 888This task is | s not applicable for me. | |

65

| SS | | | RTOG Study 0830 | Case # |
|---|---|---|---|---|
| | | | PLACE LAB | EL HERE |
| | | | Institution | Institution No. |
| | | | Participant's Initials | Partiolpant's I.D. No. |
| | 13) Kneeling is: | | | |
| | roy raisening is: | 1impossible | to do. | |
| | | 2extremely | | |
| | | 3moderately | | |
| | | 4a little bit d | ifficult. | |
| | | 5not at all di | ifficult. | |
| | | 888This task i | s not applicable for me. | |
| | 14) Bending to pick someth | | | |
| | | 1impossible | | |
| | | 2extremely | | |
| | | 3moderately<br>4a little bit d | | |
| | | 5not at all di | | |
| | | 888This task i | is not applicable for me. | |
| | 15) Walking upstairs is: | | | |
| | | 1impossible | | |
| | | 2extremely | | |
| | | 3moderately | | |
| | | 4a little bit d | | |
| | | 6not at all di | moult. | |
| | | 888This task i | is not applicable for me. | |
| | 16) Walking downstairs is: | | | |
| | | 1impossible | to do. | |
| | | 2extremely | difficult. | |
| | | 3moderately | y difficult. | |
| | | 4a little bit d | ifficult. | |
| | | 5not at all di | ifficult. | |
| | | 888This task i | s not applicable for me. | |
| ( | | | | |

| 99 | RTOG Study 0830 | Case # |
|---|---|---|
| | PLAC | E LABEL HERE |
| | Institution | |
| | Participant's Initials | Institution No. Partiolpant's I.D. No. |
| at the leading to | | |
| 17) Driving Is: | impossible to de | |
| 1 2 | | |
| 3 | | |
| 4 | | |
| 5 | | |
| 886 | This task is not applicable for me | |
| 18) Walking within the house is | | |
| 1 | | |
| 2 | | |
| | moderately difficult. | |
| | a little bit difficult.<br>not at all difficult. | |
| | not at all dillicult. | |
| 886 | This task is not applicable for me | |
| 9) Walking outdoors is: | | |
| 1 | impossible to do. | |
| 2 | extremely difficult. | |
| 3 | moderately difficult. | |
| 4 | a little bit difficult. | |
| 5 | not at all difficult. | |
| 888 | This task is not applicable for me | |
| 20) Sitting Is: | | |
| | impossible to do. | |
| | extremely difficult. | |
| | moderately difficult. | |
| | a little bit difficult. | |
| 5 | not at all difficult. | |
| 886 | This task is not applicable for me | |

| SS | | RTOG Study 0830 | Case #<br>ABEL HERE |
|---|---|---|---|
| | | Institution Participant's Initials | Institution No. Participant's I.D. No. |
| 21) Walking up or down hills | or a ramp is: | | |
| | 1Impossible to | do. | |
| | 2extremely diff | lcuit. | |
| | 3moderately di | moult. | |
| | 4a little bit diffic | cult. | |
| | 6not at all diffic | sult. | |
| | 888This task is n | ot applicable for me. | |
| 22) Standing upright is: | | | |
| | 1Impossible to | do. | |
| | 2extremely diff | | |
| | 3moderately di | | |
| | 4a little bit diffic | | |
| | 5not at all diffic | sult. | |
| | 888This task is n | ot applicable for me. | |
| 23) Getting up from kneeling | ls: | | |
| | 1Impossible to | do. | |
| | 2extremely diff | louit. | |
| | 3moderately di | fficult. | |
| | 4a little bit diffic | cult. | |
| | 5not at all diffic | sult. | |
| | 888This task is n | ot applicable for me. | |
| 24) Getting in and out of a ca | rls: | | |
| | 1Impossible to | | |
| | 2extremely diff | louit. | |
| | 3moderately di | ffcult. | |
| | 4a little bit diffic | | |
| | 5not at all diffic | suit. | |
| | 888This task is n | ot applicable for me. | |

| 00 | | RTOG Study 0830 | Case # |
|---|---|---|---|
| 33 | | | |
| | | PLACE LAB | EL HERE |
| | | Institution | Institution No. |
| | | Participant's Initials | Participant's I.D. No. |
| | 25) Participating in sexual activities is: | | |
| | 1impossible to do. | | |
| | 2extremely difficult. | | |
| | 3moderately difficult | L. | |
| | 4 a little bit difficult. | | |
| | 5 not at all difficult. | | |
| | 888This task is not ap | plicable for me. | |
| | 26) Completing my usual duties at work is: (Work inclu | ides both a job outside the home a | and as a homemaker.) |
| | 1impossible to do. | | , |
| | 2extremely difficult. | | |
| | 3moderately difficult | t. | |
| | 4a little bit difficult. | | |
| | 5not at all difficult. | | |
| | 888This task is not ap 27) Working my usual number of hours is: (Work | | the home and as a |
| | homemaker.) | | |
| | 1impossible to do. | | |
| | 2extremely difficult. | | |
| | 3moderately difficult | t. | |
| | 4a little bit difficult. | | |
| | 5not at all difficult. | | |
| | 888This task is not ap | oplicable for me. | |
| | 28) Participating in my usual leisure activities is: | | |
| | 1impossible to do. | | |
| | 2extremely difficult. | | |
| | 3moderately difficult | t. | |
| | 4a little bit difficult. | | |
| | 5not at all difficult. | | |
| | 888This task is not ap | plicable for me. | |

MC1973

| | | RTOG Study 0830 | Case # |
|---|---|---|---|
| | | PLACI | E LABEL HERE |
| | | Institution | Institution No. |
| | | Participant's initials | Partiolpant's I. |
| 29) Socializing with friends and fami | ilv is: | | |
| | impossible to do. | | |
| | extremely difficult. | | |
| | moderately difficult. | | |
| 4 | a little bit difficult. | | |
| 5 | not at all difficult. | | |
| 888 | This task is not app | olicable for me. | |
| 30) Participating in my usual sportin | g activities is: | | |
| 1 | impossible to do. | | |
| 2 | extremely difficult. | | |
| 3 | moderately difficult. | | |
| | a little bit difficult. | | |
| 6 | not at all difficult. | | |
| 888 | This task is not app | olicable for me. | |
| 1) Considering all the activities in w | hich I participate i | n daily life, I would rate th | e ability to perform these |
| activities during the past week as: | | | |
| activities during the past week as: | _impossible to do. | | |
| | extremely difficult | | |
| 1 | extremely difficult<br>moderately difficu | | |
| 1<br>2<br>3<br>4 | extremely difficult<br>moderately difficult<br>a little bit difficult. | | |
| 1<br>2<br>3<br>4<br>5 | extremely difficult<br>moderately difficu | | |
| 1234 | extremely difficult<br>moderately difficult<br>a little bit difficult.<br>not at all difficult. | h. | |
| 1<br>2<br>3<br>4<br>5<br>2) I would rate myself as being : | extremely difficult<br>moderately difficult<br>a little bit difficult.<br>not at all difficult.<br>completely disable | lt. | |
| 1 | extremely difficult moderately difficult. a little bit difficult. not at all difficult. completely disable severely disabled | lt.<br>od | |
| 1 | extremely difficult moderately difficult. a little bit difficult. not at all difficult. completely disable severely disabled moderately disabled | lt.<br>od | |
| 1 | extremely difficult moderately difficult. a little bit difficult. not at all difficult. completely disable severely disabled moderately disable mildly disabled. | od<br>lod. | |
| 1 | extremely difficult moderately difficult. a little bit difficult. not at all difficult. completely disable severely disabled moderately disabled not at all disabled not at all disabled. | ed<br>lod. | |
| 1 | extremely difficult moderately difficult. a little bit difficult. not at all difficult. completely disable severely disabled moderately disable mildly disabled. not at all disabled ies you find difficult | ed . ed to perform or on any othe | |
| 2 3 4 5 2) I would rate myself as being: 1 2 3 4 5 4 5 5 5 6 6 6 6 6 6 6 6 6 6 6 6 6 6 | extremely difficult moderately difficult. a little bit difficult. not at all difficult. completely disable severely disabled moderately disable mildly disabled. not at all disabled ies you find difficult | ed . ed to perform or on any othe | |
| 1 | extremely difficult moderately difficult. a little bit difficult. not at all difficult. completely disable severely disabled moderately disable mildly disabled. not at all disabled ies you find difficult | ed . ed to perform or on any othe | |

70

# Appendix IV

# Joint Stiffness Assessment (Specific to ipsilateral extremity/region)

| MC: |
|---|
| Patient Name: |
| Date of Assessment: |
| Name of Assessor: |
| Was Joint Stiffness Present: Yes/No (circle one) |
| If yes, Joint Affected: Upper proximal extremity Upper distal extremity (includes elbow) Lower proximal extremity (includes knee) Lower distal extremity Superficial trunk |
| Grade: □ 1- Mild stiffness; slight ROM loss □ 2 - Moderate stiffness; pain, ROM loss □ 3 - Severe stiffness, pain, ROM loss □ 4 - Necrosis; complete fixation |
| Attribution to RT: Definite Possible Probable Unlikely Unrelated |
| Attribution to Surgery: Definite Possible Probable Unlikely Unrelated |

## Appendix V

# Regional Alopecia Assessment

| MC: |
|---|
| Patient Name: |
| Date of Assessment: |
| Name of Assessor: |
| Was Regional Alopecia Present: Yes/No |
| If yes, Region Affected: Upper proximal extremity Upper distal extremity (includes elbow) Lower proximal extremity (includes knee) Lower distal extremity Superficial trunk |
| Grade: □ 1 - Hair loss of <50% of normal for that individual that is not obvious on close inspection □ 2 - Hair loss of >50% normal for that individual that is readily apparent b others |
| Attribution to RT: Definite Possible Probable Unlikely Unrelated |

# Appendix VI

## **Surgical Wound Complication Assessment**

| MC: |
|-------------------------------------------------------------------------|
| Patient Name: |
| Name of Assessor: |
| Surgical wound complication: Yes/No |
| If yes, |
| Surgical wound start date: |
| Surgical wound end date: Date notified of surgical wound complication: |
| Surgical wound complication classification: |
| Wound management via secondary unplanned operation under anesthesia |
| ☐ Wound management via invasive procedures other than operation |
| Surgical wound complication procedure performed: |